CLINICAL TRIAL: NCT02657434
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab (MPDL3280A, Anti-Pd-L1 Antibody) in Combination With Carboplatin or Cisplatin + Pemetrexed Compared With Carboplatin or Cisplatin + Pemetrexed in Patients Who Are Chemotherapy-Naive and Have Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Combination With Carboplatin or Cisplatin + Pemetrexed Compared With Carboplatin or Cisplatin + Pemetrexed in Participants Who Are Chemotherapy-Naive and Have Stage IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC) (IMpower 132)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29438; 2015-003605-42 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-15 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Carboplatin; Cisplatin; Pemetrexed

ARMS (2):
- Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed (Experimental): Participants received intravenous (IV) infusion of 1200 milligrams (mg) of atezolizumab on Day 1 every 3 weeks (q3w), IV infusion of 500 milligrams per meter square (mg/m^2) pemetrexed on Day 1 q3w, and as per investigator's choice either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain area under concentration versus time (AUC) = 6 milligrams per milliliter per minute (mg/mL/min) or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period of 4 or 6 cycles (Cycle length=21 days). Participants who experienced clinical benefit during the induction phase began maintenance therapy. Participants will receive IV infusion of 1200 mg of atezolizumab and 500 mg/m^2 of pemetrexed on Day 1 q3w until disease progression in the maintenance period.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Arm B (Carboplatin or Cisplatin + Pemetrexed) (Active Comparator): Participants received IV infusion of 500 mg/m^2 pemetrexed on Day 1 q3w, and as per investigator's choice of either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain AUC =6 mg/mL/min or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period for 4 or 6 cycles (Cycle length=21 days). Participants who did not experience disease progression during the induction phase began maintenance therapy. Participants will receive IV infusion of 500 mg/m^2 of pemetrexed on Day 1 q3w until disease progression in the maintenance period.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — Participants received IV infusion of 1200 mg atezolizumab on Day 1 q3w for 4 or 6 cycles (Cycle length=21 days) in induction dosing period and until disease progression on Day 1 q3w in the maintenance dosing period.
  Other Names: MPDL3280A; TECENTRIQ
  Arms: Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Drug: Carboplatin — Participants received IV infusion of carboplatin on Day 1 q3w for 4 or 6 cycles (Cycle length=21 days) in induction dosing period with doses calculated using Calvart formula.
Drug: Cisplatin — Participants received IV infusion of 75 mg/m^2 cisplatin on Day 1 q3w for 4 or 6 cycles (Cycle length=21 days) in induction dosing period.
Drug: Pemetrexed — Participants received IV infusion of 500 mg/m^2 pemetrexed on Day 1 q3w for 4 or 6 cycles (Cycle length=21 days) in induction dosing period and until disease progression on Day 1 q3w in the maintenance dosing period.

SUMMARY:
This is a randomized, Phase III, multicenter, open-label study designed to evaluate the safety and efficacy of atezolizumab in combination with cisplatin or carboplatin + pemetrexed compared with treatment with cisplatin or carboplatin + pemetrexed in participants who are chemotherapy-naive and have Stage IV non-squamous NSCLC. Eligible participants will be randomized by a 1:1 ratio into 2 groups: Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed) and Arm B (Carboplatin or Cisplatin + Pemetrexed). The study will be conducted in two phases: Induction Phase and Maintenance Phase.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed, Stage IV non-squamous NSCLC. Participants with tumors of mixed non-small cell histology (i.e., squamous and non-squamous) are eligible if the major histological component appears to be non-squamous
* No prior treatment for Stage IV non-squamous NSCLC. Participants with a sensitizing mutation in the epidermal growth factor receptor (EGFR) gene or with an anaplastic lymphoma kinase (ALK) fusion oncogene are excluded. Participants with unknown EGFR and ALK status require test results at screening from a local or central laboratory
* Participants who have received prior neo-adjuvant, radiotherapy, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from randomization since the last dose of chemotherapy and/or radiotherapy
* Participants should submit a pre-treatment tumor tissue sample if available before or within 4 weeks after enrollment. If tumor tissue is not available, participants are still eligible
* For participants enrolled in the extended China enrollment phase: current resident of mainland China, Hong Kong, or Taiwan and of Chinese ancestry
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 5 months after the last dose of atezolizumab or 6 months after the last dose of cisplatin
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

Cancer-Specific Exclusions

* Participants with a sensitizing mutation in the EGFR gene or an ALK fusion oncogene
* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for greater than or equal to (>= 2) weeks prior to randomization
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia (greater than [>] 1.5 millimole/Liter ionized calcium or calcium >12 milligrams/deciliter or corrected serum calcium >upper limit of normal)
* Malignancies other than NSCLC within 5 years prior to randomization
* Known tumor programmed death-ligand 1 (PD-L1) expression status from other clinical studies (e.g., participants whose PD-L1 expression status was determined during screening for entry into a study with anti-PD-1 or anti-PD L1 antibodies but were not eligible are excluded)

General Medical Exclusions:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of certain autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis
* All participants will be tested for human immunodeficiency virus (HIV) prior to the inclusion into the study and HIV-positive participants will be excluded from the clinical study
* Severe infections within 4 weeks prior to randomization
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to randomization, unstable arrhythmias, or unstable angina
* Illness or condition that may interfere with a participant's capacity to understand, follow, and/or comply with study procedures

Exclusion Criteria Related to Medications and Chemotherapy:

* Prior treatment with EGFR inhibitors or ALK inhibitors
* Any approved anti-cancer therapy, including hormonal therapy within 21 days prior to initiation of study treatment
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks prior to randomization
* Treatment with systemic immunosuppressive medications

Exclusion Criteria Related to Chemotherapy:

* History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds
* Participants with hearing impairment (cisplatin)
* Grade >=2 peripheral neuropathy as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria (cisplatin)
* Creatinine clearance (CRCL) <60 milliliters/minute (mL/min) for cisplatin or <45 mL/min for carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (183):
- United States (26):
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - St. Joseph Heritage Healthcare, Sebastopol, California
  - Stamford Hospital; BCC, MOHR, Stamford, Connecticut
  - Orlando Health Inc., Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Northside Hospital, Atlanta, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - HealthCare Research Network II, LLC - PPDS, Tinley Park, Illinois
  - Fort Wayne Med Oncology & Hematology Inc, Fort Wayne, Indiana
  - Goshen Health System, Goshen, Indiana
  - University of Kentucky; Markey Cancer Center, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - CHI Health St. Francis, Grand Island, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Swedish Cancer Institute, Cary, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Oncology Consultants PA, Houston, Texas
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - St. Vincent Hospital, Green Bay, Wisconsin
- Argentina (3):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires
  - Fundacion Clinica Colombo, Córdoba
  - Clinica Viedma S.A., Viedma
- Australia (9):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Sydney Adventist Hospital; Clinical Trial Unit, Sydney, New South Wales
  - St George Hospital; Medical Oncology, Sydney, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Health Services, Ballarat, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Barwon Health, Geelong, Victoria
- Klinikum Wels-Grieskirchen GmbH, Wels, Austria
- Belgium (3):
  - AZ Maria Middelares, Ghent
  - Clinique André Renard; Pneumologie, Herstal
  - AZ Delta (Campus Rumbeke), Apotheek, Roeselare
- Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia, Bulgaria
- Chile (3):
  - Health & Care SPA, Santiago
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
  - Hospital Clinico Vina del Mar?, Viña del Mar
- China (19):
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Changzhou First People's Hospital, Changzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Anhui Provincial Hospital; 2F,Tumor chemotherapy Department, Hefei
  - Anhui Provincial Hospital; Respiratory Department, Hefei
  - Qilu Hospital, Jinan
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Tumor Center,Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Zhejiang Cancer Hospital, Zhejiang
- France (10):
  - Institut Sainte Catherine, Avignon
  - Hopital Louis Pradel; Pneumologie, Bron
  - Centre Jean Perrin Centre Regional de Lutte Contre Le Cancer D auvergne, Clermont-Ferrand
  - Centre Hospitalier Intercommunal; Service de Pneumologie, Créteil
  - Polyclinique de Limoges - Site Chenieux; Oncologie Medicale, Limoges
  - Hopital Nord AP-HM, Marseille
  - Centre Regional de Lutte contre le Cancer Val d Aurelle - Paul Lamarque; Service d oncologie, Montpellier
  - Centre Hospitalier de Mulhouse - Hopital Emile Muller, Mulhouse
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Hopital d Instruction des Armees de Sainte Anne, Toulon
- Hungary (5):
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Markusovszky Hospital, Szombathely
  - Tudogyogyintezet Torokbalint, Törökbálint
- Ireland (2):
  - Mater Misecordiae University Hospital, Dublin
  - St James's Hospital, Dublin
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Edith Wolfson Medical Center, Holon
  - Rabin Medical Center, Petach Tiqwa
- Italy (9):
  - Presidio Ospedaliero Vito Fazzi; Unita Operativa Di Oncologia Medica, Lecce, Apulia
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Ospedale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - Azienda Policlinico Umberto I, Rome, Lazio
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga; S.C.D.U. di Oncologia Toracica, Orbassano (TO), Piedmont
  - Ospedale San Vincenzo Taormina :Divisione di Oncologia Medica, Taormina, Sicily
  - Ospedale San Luca - USL2 Lucca, Lucca, Tuscany
- Japan (20):
  - National Hospital Organization Nagoya Medical Center, Aichi
  - National Cancer Center Hospital East, Chiba
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Asahikawa Medical Center, Hokkaido
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Kagoshima University Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tohoku University Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka University Hospital, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Saga University Hospital, Saga
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - NTT Medical Center Tokyo, Tokyo
  - National Hospital Organization Yamaguchi - Ube Medical Center, Yamaguchi
- Riga East Clinical University Hospital Latvian Oncology Centre, Riga, Latvia
- Panevezys Hospital, Panevezys, Lithuania
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Advanced Medical and Dental Institute; Kompleks Klinikal, Kepala Batas, Pulau Pinang
- Netherlands (6):
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis Gelderse Vallei, Ede
  - Ziekenhuis St. Jansdal, Harderwijk
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - Haga Ziekenhuis, The Hague
  - ETZ TweeSteden, Tilburg
- Hospital Nacional Cayetano Heredia, Lima, Peru
- Portugal (3):
  - Hospital Beatriz Angelo, Loures
  - Unidade Local de Saude de Matosinhos SA, Matosinhos Municipality
  - Hospital CUF Porto; Servico de Imunoalergologia, Senhora Da Hora - Porto
- Romania (3):
  - Medisprof SRL, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Constanta, Constanța
  - Euroclinic Center of Oncology SRL, Iași
- Russia (3):
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk, Moscow Oblast
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (24):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - ICO L'Hospitalet; Servicio de oncologia medica, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital de Mataro, Mataro, Cantabria
  - Onkologikoa; Ensayos Clinicos, Donostia / San Sebastian, Guipuzcoa
  - Centro Oncologico de Galicia COG; Medical Oncology, A Coruña, LA Coruña
  - Hospital Universitario Virgen de La Arrixaca; Servicio De Oncologia, El Palmar, Murcia
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Complejo Hospitalario de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Complejo Hospitalario Nuestra Senora de Valme, Seville, Sevilla
  - Hospital General Univ. de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud; Servicio de Oncologia Medica, Barcelona
  - C.A.U de Burgos- Hospital Universitario de Burgos; Servicio de Oncologia, Burgos
  - Hospital Universitari de Girona Dr Josep Trueta; Departamento de Oncologia Medica, Girona
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - HM Sanchinarro ? CIOCC, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General; Servicio de Neurologia, Málaga
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (6):
  - Buddhist Dalin Tzuchi General Hospital, Dalin, Chiayi
  - E-DA Hospital; Chest, Kaohsiung City
  - Chi Mei Medical Center Liou Ying Campus, Liuying Township
  - National Taiwan Uni Hospital; Internal Medicine, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Ukraine (6):
  - MI Dnipropetrovsk City Multifield Clinical Hospital 4 of Dnipropetrovsk Regional Council, Dnipropetrovsk, Katerynoslav Governorate
  - Kyiv Railway Clinical Hospital #3 of Branch Health Center of PJSC Ukrainian Railway; Surgery Dept, Kyiv, Kharkiv Governorate
  - MICR Oncology Dispensary of Cherkasy Regional Council; Regional Center of Clinical Oncology, Cherkasy
  - Private Enterprise Private Manufacturing Company Acinus, Kirovograd
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary; Oncothoracic department, Sumy
  - MI Zaporizhzhia Regional Clinical Oncological Dispensary Zaporizhzhia SMU Ch of Oncology, Zaporizhzhya
- United Kingdom (10):
  - Bristol Haematology and Oncology centre, Bristol
  - Velindre Hospital, Cardiff
  - Gartnavel General Hospital; Beatson West of Scotland Cancer Centre, Glasgow
  - Raigmore Hospital, Inverness
  - St George?s Hospital, London
  - Charing Cross Hospital, London
  - Churchill Hospital, Oxford
  - Derriford Hospital; Plymouth Oncology Centre, Plymouth
  - Queen's Hospital, Romford
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Socinski MA, Jotte RM, Cappuzzo F, Nishio M, Mok TSK, Reck M, Finley GG, Kaul MD, Yu W, Paranthaman N, Bara I, West HJ. Association of Immune-Related Adverse Events With Efficacy of Atezolizumab in Patients With Non-Small Cell Lung Cancer: Pooled Analyses of the Phase 3 IMpower130, IMpower132, and IMpower150 Randomized Clinical Trials. JAMA Oncol. 2023 Apr 1;9(4):527-535. doi: 10.1001/jamaoncol.2022.7711. PMID 36795388
- [Derived] Lu S, Fang J, Wang Z, Fan Y, Liu Y, He J, Zhou J, Hu J, Xia J, Liu W, Shi J, Yi J, Cao L. Results from the IMpower132 China cohort: Atezolizumab plus platinum-based chemotherapy in advanced non-small cell lung cancer. Cancer Med. 2023 Feb;12(3):2666-2676. doi: 10.1002/cam4.5144. Epub 2022 Sep 2. PMID 36052772
- [Derived] Ton TGN, Pal N, Trinh H, Mahrus S, Bretscher MT, Machado RJM, Sadetsky N, Chaudhary N, Lu MW, Riely GJ. Replication of Overall Survival, Progression-Free Survival, and Overall Response in Chemotherapy Arms of Non-Small Cell Lung Cancer Trials Using Real-World Data. Clin Cancer Res. 2022 Jul 1;28(13):2844-2853. doi: 10.1158/1078-0432.CCR-22-0471. PMID 35511917

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is considered "Completed" because the planned study activities and analyses have been performed.
Period: Overall Study
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Started | 286 | 292
Completed | 0 | 0
Not Completed | 286 | 292
Not completed — Study Terminated By Sponsor | 64 | 82
Not completed — Death | 189 | 190
Not completed — Lost to Follow-up | 2 | 2
Not completed — Randomization by Error | 2 | 0
Not completed — Withdrawal by Subject | 28 | 17
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm B (Carboplatin or Cisplatin + Pemetrexed): Participants received IV infusion of 500 mg/m^2 pemetrexed on Day 1 q3w, and as per investigator's choice of either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain AUC =6 mg/mL/min or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period for 4 or 6 cycles (Cycle length=21 days). Participants who did not experience disease progression during the induction phase will begin maintenance therapy. Participants will receive IV infusion of 500 mg/m^2 of pemetrexed on Day 1 q3w until disease progression in the maintenance period.
- Total: Total of all reporting groups
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed | Total
Number analyzed (Participants) | 286 | 292 | 578
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (9.4) | 63.3 (9.4) | 62.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 100 | 194
  Male | 192 | 192 | 384
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 17 | 38
  Not Hispanic or Latino | 241 | 243 | 484
  Unknown or Not Reported | 24 | 32 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 65 | 71 | 136
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 203 | 193 | 396
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 25 | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator using RECIST v1.1 or death from any cause, whichever occurred first.
Time Frame: Randomization up to approximately 39 months
Population: The ITT population was defined as all randomized patients, whether or not the patients received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Months | 5.2 [4.3 to 5.6] | 7.7 [6.7 to 8.5]
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Other — Unstratified Analysis; p < 0.0001, Log Rank; Hazard Ratio, log = 0.562, 95% CI 2-sided [0.471 to 0.671]

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomization to death from any cause.
Time Frame: Randomization up to approximately 39 months
Population: The ITT population was defined as all randomized patients, whether or not the patients received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Months | 13.6 [11.0 to 15.7] | 17.5 [13.2 to 19.6]
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority — Unstratified Analysis; p = 0.1559, Log Rank; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.709 to 1.056]
Statistical Analysis 2: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority — Stratified Analysis; p = 0.1546, Log Rank; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.707 to 1.056]

3. Secondary Outcome: Overall Survival Rate at Year 1
Description: The Overall Survival Rate at the 1-year landmark time point is defined as the probabilities that participants are alive 1-year after randomization.
Time Frame: Year 1
Population: The ITT population was defined as all randomized patients, whether or not the patients received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Percentage | 55.04 [49.21 to 60.87] | 59.72 [54.02 to 65.41]
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority; p = 0.2606, z test; Difference in event free rate = 4.68, 95% CI 2-sided [-3.47 to 12.83]

4. Secondary Outcome: Overall Survival Rate Year 2
Description: The Overall Survival Rate at the 2-year landmark time point is defined as the probabilities that participants are alive 2-years after randomization.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Percentage | 34.01 [28.40 to 39.62] | 39.13 [33.44 to 44.81]
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority; p = 0.2090, Z-test; Difference in Event Free Rate = 5.12, 95% CI 2-sided [-2.87 to 13.11]

5. Secondary Outcome: Percentage of Participants With an Objective Response (Complete Response [CR] or Partial Response [PR]) Assessed by the Investigator Using RECIST V1.1
Description: An objective response is defined as either an unconfirmed CR or a PR, as determined by the investigator using RECIST v1.1. Objective Response Rate is defined as the proportion of patients who had an objective response.
Time Frame: Randomization up to approximately 25 months
Population: The ITT population was defined as all randomized patients, whether or not the patients received the assigned treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Percentage of Participants
  Responders | 37.4 | 51.7
  Non-Responders | 62.6 | 48.3
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Difference in response rate = 14.3, 95% CI 2-sided [5.9 to 22.7]

6. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using RECIST v1.1
Description: DOR is defined as the time interval from the date of the first occurrence of a CR or PR (whichever status is recorded first) until the first date that progressive disease or death is documented, whichever occurs first.
Time Frame: Randomization up to approximately 25 months
Population: DOR was assessed in participants who had an objective response as determined by the investigator using RECIST v1.1.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 286 | 292
Months | 6.4 [4.4 to 7.6] | 9.5 [6.9 to 12.2]
Statistical Analysis 1: Comparison: Arm B (Carboplatin or Cisplatin + Pemetrexed) vs Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed; Test type: Superiority; p = 0.0024, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.85]

7. Secondary Outcome: Change From Baseline in Patient-Reported Lung Cancer Symptoms as Assessed by European Organization for the Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire-Core 30 (QLQ-C30) Symptom Score
Description: EORTC QLQ-C30 is a validated and reliable self-report measure that consists of 30 questions that assess five aspects of patient functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), global health/quality of life, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). EORTC QLQ-C30 is scored according to the EORTC scoring manual (Fayers et al. 2001). All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high or healthy level of functioning/HRQoL (Health-Related Quality of Life); however a high score for a symptom scale or item represents a high level of symptomatology or problems. A ≥10-point change in the symptoms subscale score is perceived by patients as clinically significant (Osoba et al. 1998).
Time Frame: Baseline up to 3 and 6 months after disease progression or loss of clinical benefit (up to approximately 25 months)
Population: ITT population with a non-missing baseline and at least a post-baseline PRO assessment (i.e., PRO evaluable population).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 232 | 242
Units on a scale
  Dyspnoea: Week 3: number analyzed (Participants) | 222 | 216
  Dyspnoea: Week 3 | -1.95 (23.97) | -1.39 (25.17)
  Dyspnoea: Week 6: number analyzed (Participants) | 189 | 198
  Dyspnoea: Week 6 | -1.23 (23.16) | -4.71 (26.66)
  Dyspnoea: Week 9: number analyzed (Participants) | 166 | 179
  Dyspnoea: Week 9 | 0.20 (26.34) | -6.33 (26.62)
  Dyspnoea: Week 12: number analyzed (Participants) | 147 | 177
  Dyspnoea: Week 12 | -0.91 (27.57) | -3.39 (29.10)
  Dyspnoea: Week 15: number analyzed (Participants) | 140 | 164
  Dyspnoea: Week 15 | -1.67 (28.92) | -2.44 (28.73)
  Dyspnoea: Week 18: number analyzed (Participants) | 126 | 155
  Dyspnoea: Week 18 | -2.12 (24.85) | -3.44 (30.43)
  Dyspnoea: Week 21: number analyzed (Participants) | 100 | 150
  Dyspnoea: Week 21 | -5.67 (29.61) | -2.89 (31.83)
  Dyspnoea: Week 24: number analyzed (Participants) | 97 | 136
  Dyspnoea: Week 24 | -2.75 (28.74) | -2.45 (31.85)
  Dyspnoea: Week 27: number analyzed (Participants) | 79 | 126
  Dyspnoea: Week 27 | -2.53 (31.47) | -1.32 (27.13)
  Dyspnoea: Week 30: number analyzed (Participants) | 80 | 123
  Dyspnoea: Week 30 | -1.25 (32.45) | -2.71 (28.50)
  Dyspnoea: Week 33: number analyzed (Participants) | 73 | 107
  Dyspnoea: Week 33 | -1.83 (27.15) | -3.74 (30.14)
  Dyspnoea: Week 36: number analyzed (Participants) | 61 | 105
  Dyspnoea: Week 36 | -3.83 (30.49) | -6.67 (31.49)
  Dyspnoea: Week 39: number analyzed (Participants) | 60 | 95
  Dyspnoea: Week 39 | -1.67 (31.55) | -8.42 (29.16)
  Dyspnoea: Week 42: number analyzed (Participants) | 51 | 95
  Dyspnoea: Week 42 | -3.27 (28.48) | -9.12 (28.12)
  Dyspnoea: Week 45: number analyzed (Participants) | 48 | 79
  Dyspnoea: Week 45 | -6.25 (32.00) | -2.11 (30.82)
  Dyspnoea: Week 48: number analyzed (Participants) | 39 | 81
  Dyspnoea: Week 48 | -5.13 (32.03) | -7.41 (26.87)
  Dyspnoea: Week 51: number analyzed (Participants) | 36 | 80
  Dyspnoea: Week 51 | -14.81 (30.28) | -2.92 (26.09)
  Dyspnoea: Week 54: number analyzed (Participants) | 31 | 72
  Dyspnoea: Week 54 | -9.68 (35.69) | -2.78 (27.26)
  Dyspnoea: Week 57: number analyzed (Participants) | 26 | 71
  Dyspnoea: Week 57 | -7.69 (28.76) | -5.63 (28.72)
  Dyspnoea: Week 60: number analyzed (Participants) | 18 | 56
  Dyspnoea: Week 60 | -11.11 (25.57) | 0.00 (25.43)
  Dyspnoea: Week 63: number analyzed (Participants) | 13 | 39
  Dyspnoea: Week 63 | -7.69 (14.62) | -5.13 (23.62)
  Dyspnoea: Week 66: number analyzed (Participants) | 7 | 37
  Dyspnoea: Week 66 | -9.52 (16.27) | -1.80 (24.78)
  Dyspnoea: Week 69: number analyzed (Participants) | 6 | 28
  Dyspnoea: Week 69 | -16.67 (18.26) | -3.57 (24.58)
  Dyspnoea: Week 72: number analyzed (Participants) | 8 | 22
  Dyspnoea: Week 72 | -4.17 (27.82) | 0.00 (27.22)
  Dyspnoea: Week 75: number analyzed (Participants) | 5 | 23
  Dyspnoea: Week 75 | -6.67 (14.91) | -5.80 (19.21)
  Dyspnoea: Week 78: number analyzed (Participants) | 2 | 14
  Dyspnoea: Week 78 | 0.00 (0.00) | -4.76 (25.68)
  Dyspnoea: Week 81: number analyzed (Participants) | 2 | 9
  Dyspnoea: Week 81 | 0.00 (0.00) | -11.11 (23.57)
  Dyspnoea: Week 84: number analyzed (Participants) | 2 | 8
  Dyspnoea: Week 84 | 0.00 (0.00) | -4.17 (21.36)
  Dyspnoea: Week 87: number analyzed (Participants) | 1 | 4
  Dyspnoea: Week 87 | 0.00 (NA) — Only 1 participant. | 8.33 (16.67)
  Dyspnoea: Week 90: number analyzed (Participants) | 1 | 2
  Dyspnoea: Week 90 | 0.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Dyspnoea: Week 93: number analyzed (Participants) | 0 | 1
  Dyspnoea: Week 93 |  | 0.00 (NA) — Only 1 participant.
  Dyspnoea: Time of First Pd: number analyzed (Participants) | 0 | 0
  Dyspnoea: Time of Last Tx Dose: number analyzed (Participants) | 0 | 0
  Dyspnoea: Survival Follow-Up Week 12: number analyzed (Participants) | 29 | 25
  Dyspnoea: Survival Follow-Up Week 12 | 9.20 (35.52) | 8.00 (42.25)
  Dyspnoea: Survival Follow-Up Week 24: number analyzed (Participants) | 19 | 7
  Dyspnoea: Survival Follow-Up Week 24 | 5.26 (25.49) | -14.29 (17.82)

8. Secondary Outcome: Change From Baseline in Patient-Reported Lung Cancer Symptoms as Assessed by EORTC Quality-of-Life Lung Cancer Module (QLQ-LC13) Symptom Score
Description: The EORTC QLQ-LC13 module incorporates one multiple item scale to assess dyspnea and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. The EORTC QLQ-LC13 is scored according to the EORTC scoring manual (Fayers et al. 2001). All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high or healthy level of functioning/HRQoL (Health-Related Quality of Life); however, a high score for a symptom scale or item represents a high level of symptomatology or problems. A≥10-point change in the symptoms subscale score is perceived by patients as clinically significant (Osoba et al. 1998).
Time Frame: Baseline up to 3 and 6 months after disease progression or loss of clinical benefit (up to approximately 25 months)
Population: ITT population with a non-missing baseline and at least a post-baseline PRO assessment (i.e., PRO evaluable population).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 230 | 234
Units on a scale
  Coughing: Week 3: number analyzed (Participants) | 213 | 205
  Coughing: Week 3 | -2.50 (25.37) | -3.41 (26.90)
  Coughing: Week 6: number analyzed (Participants) | 187 | 190
  Coughing: Week 6 | -3.57 (27.20) | -9.82 (26.50)
  Coughing: Week 9: number analyzed (Participants) | 162 | 173
  Coughing: Week 9 | -1.85 (24.43) | -8.29 (31.37)
  Coughing: Week 12: number analyzed (Participants) | 145 | 168
  Coughing: Week 12 | -3.91 (28.46) | -10.71 (31.66)
  Coughing: Week 15: number analyzed (Participants) | 137 | 159
  Coughing: Week 15 | -6.33 (30.39) | -11.53 (29.05)
  Coughing: Week 18: number analyzed (Participants) | 125 | 149
  Coughing: Week 18 | -4.00 (26.97) | -11.63 (27.92)
  Coughing: Week 21: number analyzed (Participants) | 100 | 146
  Coughing: Week 21 | -6.00 (27.78) | -10.50 (30.76)
  Coughing: Week 24: number analyzed (Participants) | 97 | 133
  Coughing: Week 24 | -4.81 (28.05) | -10.03 (33.08)
  Coughing: Week 27: number analyzed (Participants) | 78 | 123
  Coughing: Week 27 | -3.85 (26.85) | -11.65 (34.40)
  Coughing: Week 30: number analyzed (Participants) | 80 | 120
  Coughing: Week 30 | 0.42 (29.76) | -11.39 (31.31)
  Coughing: Week 33: number analyzed (Participants) | 72 | 103
  Coughing: Week 33 | -0.46 (26.53) | -11.97 (30.91)
  Coughing: Week 36: number analyzed (Participants) | 60 | 103
  Coughing: Week 36 | -6.11 (31.59) | -12.94 (30.33)
  Coughing: Week 39: number analyzed (Participants) | 60 | 92
  Coughing: Week 39 | -5.00 (30.58) | -13.41 (32.43)
  Coughing: Week 42: number analyzed (Participants) | 52 | 93
  Coughing: Week 42 | -8.97 (27.31) | -14.70 (29.68)
  Coughing: Week 45: number analyzed (Participants) | 48 | 77
  Coughing: Week 45 | -13.19 (28.13) | -14.72 (27.83)
  Coughing: Week 48: number analyzed (Participants) | 39 | 79
  Coughing: Week 48 | -7.69 (31.96) | -13.92 (32.29)
  Coughing: Week 51: number analyzed (Participants) | 36 | 79
  Coughing: Week 51 | -17.59 (25.80) | -10.97 (34.48)
  Coughing: Week 54: number analyzed (Participants) | 31 | 70
  Coughing: Week 54 | -17.20 (27.04) | -13.81 (33.81)
  Coughing: Week 57: number analyzed (Participants) | 26 | 69
  Coughing: Week 57 | -11.54 (22.98) | -13.53 (29.33)
  Coughing: Week 60: number analyzed (Participants) | 19 | 56
  Coughing: Week 60 | -14.04 (27.92) | -10.71 (31.21)
  Coughing: Week 63: number analyzed (Participants) | 13 | 39
  Coughing: Week 63 | -10.26 (21.01) | -12.82 (27.16)
  Coughing: Week 66: number analyzed (Participants) | 7 | 37
  Coughing: Week 66 | -9.52 (25.20) | -12.61 (28.71)
  Coughing: Week 69: number analyzed (Participants) | 6 | 28
  Coughing: Week 69 | -11.11 (27.22) | -11.90 (30.38)
  Coughing: Week 72: number analyzed (Participants) | 8 | 22
  Coughing: Week 72 | -8.33 (23.57) | -16.67 (30.43)
  Coughing: Week 75: number analyzed (Participants) | 5 | 23
  Coughing: Week 75 | -13.33 (18.26) | -18.84 (28.12)
  Coughing: Week 78: number analyzed (Participants) | 2 | 14
  Coughing: Week 78 | -16.67 (23.57) | -23.81 (27.51)
  Coughing: Week 81: number analyzed (Participants) | 2 | 9
  Coughing: Week 81 | -16.67 (23.57) | -18.52 (33.79)
  Coughing: Week 84: number analyzed (Participants) | 2 | 8
  Coughing: Week 84 | -33.33 (0.00) | -29.17 (27.82)
  Coughing: Week 87: number analyzed (Participants) | 1 | 4
  Coughing: Week 87 | 0.00 (NA) — Only 1 participant. | -25.00 (31.91)
  Coughing: Week 90: number analyzed (Participants) | 1 | 2
  Coughing: Week 90 | -33.33 (NA) — Only 1 participant. | -16.67 (23.57)
  Coughing: Week 93: number analyzed (Participants) | 0 | 1
  Coughing: Week 93 |  | 0.00 (NA) — Only 1 participant.
  Coughing: Time of First Pd: number analyzed (Participants) | 61 | 70
  Coughing: Time of First Pd | -6.01 (30.13) | -10.48 (28.68)
  Coughing: Time of Last Tx Dose: number analyzed (Participants) | 199 | 201
  Coughing: Time of Last Tx Dose | -5.19 (28.05) | -8.13 (28.78)
  Coughing: Survival Follow-Up Week 12: number analyzed (Participants) | 28 | 24
  Coughing: Survival Follow-Up Week 12 | 3.57 (29.17) | -6.94 (34.02)
  Coughing: Survival Follow-Up Week 24: number analyzed (Participants) | 19 | 7
  Coughing: Survival Follow-Up Week 24 | -8.77 (24.45) | -14.29 (32.53)
  Dyspnoea: Week 3: number analyzed (Participants) | 213 | 205
  Dyspnoea: Week 3 | 0.21 (18.69) | -1.41 (17.68)
  Dyspnoea: Week 6: number analyzed (Participants) | 187 | 190
  Dyspnoea: Week 6 | 0.12 (17.13) | -1.17 (18.85)
  Dyspnoea: Week 9: number analyzed (Participants) | 162 | 173
  Dyspnoea: Week 9 | 0.89 (20.68) | -3.34 (18.65)
  Dyspnoea: Week 12: number analyzed (Participants) | 145 | 168
  Dyspnoea: Week 12 | 1.15 (21.82) | -0.46 (21.76)
  Dyspnoea: Week 15: number analyzed (Participants) | 137 | 159
  Dyspnoea: Week 15 | 0.00 (21.30) | -1.12 (20.78)
  Dyspnoea: Week 18: number analyzed (Participants) | 125 | 149
  Dyspnoea: Week 18 | -1.07 (18.90) | -3.88 (21.92)
  Dyspnoea: Week 21: number analyzed (Participants) | 100 | 146
  Dyspnoea: Week 21 | -3.56 (22.77) | -1.45 (21.85)
  Dyspnoea: Week 24: number analyzed (Participants) | 97 | 133
  Dyspnoea: Week 24 | -2.29 (21.75) | -0.42 (23.82)
  Dyspnoea: Week 27: number analyzed (Participants) | 78 | 123
  Dyspnoea: Week 27 | -0.71 (22.32) | -2.08 (19.83)
  Dyspnoea: Week 30: number analyzed (Participants) | 80 | 120
  Dyspnoea: Week 30 | 1.25 (22.57) | -2.78 (20.33)
  Dyspnoea: Week 33: number analyzed (Participants) | 72 | 103
  Dyspnoea: Week 33 | 0.77 (21.45) | -3.02 (22.82)
  Dyspnoea: Week 36: number analyzed (Participants) | 60 | 103
  Dyspnoea: Week 36 | -1.11 (20.93) | -2.91 (23.70)
  Dyspnoea: Week 39: number analyzed (Participants) | 60 | 92
  Dyspnoea: Week 39 | 1.30 (26.91) | -4.95 (22.31)
  Dyspnoea: Week 42: number analyzed (Participants) | 52 | 93
  Dyspnoea: Week 42 | -0.43 (22.65) | -6.33 (18.64)
  Dyspnoea: Week 45: number analyzed (Participants) | 48 | 77
  Dyspnoea: Week 45 | -2.08 (26.60) | -3.61 (21.36)
  Dyspnoea: Week 48: number analyzed (Participants) | 39 | 79
  Dyspnoea: Week 48 | -4.56 (24.94) | -5.34 (21.49)
  Dyspnoea: Week 51: number analyzed (Participants) | 36 | 79
  Dyspnoea: Week 51 | -9.88 (21.87) | -1.69 (18.41)
  Dyspnoea: Week 54: number analyzed (Participants) | 31 | 70
  Dyspnoea: Week 54 | -6.45 (24.47) | -1.90 (19.10)
  Dyspnoea: Week 57: number analyzed (Participants) | 26 | 69
  Dyspnoea: Week 57 | -2.99 (23.42) | -4.99 (22.99)
  Dyspnoea: Week 60: number analyzed (Participants) | 19 | 56
  Dyspnoea: Week 60 | -11.11 (23.42) | -0.40 (22.32)
  Dyspnoea: Week 63: number analyzed (Participants) | 13 | 39
  Dyspnoea: Week 63 | -6.84 (15.41) | -6.55 (23.04)
  Dyspnoea: Week 66: number analyzed (Participants) | 7 | 37
  Dyspnoea: Week 66 | -9.52 (16.27) | -4.50 (21.98)
  Dyspnoea: Week 69: number analyzed (Participants) | 6 | 28
  Dyspnoea: Week 69 | -16.67 (21.94) | -4.76 (23.12)
  Dyspnoea: Week 72: number analyzed (Participants) | 8 | 22
  Dyspnoea: Week 72 | -5.56 (19.70) | -1.52 (24.56)
  Dyspnoea: Week 75: number analyzed (Participants) | 5 | 23
  Dyspnoea: Week 75 | -6.67 (14.91) | -6.76 (17.64)
  Dyspnoea: Week 78: number analyzed (Participants) | 2 | 14
  Dyspnoea: Week 78 | 0.00 (0.00) | -3.17 (21.09)
  Dyspnoea: Week 81: number analyzed (Participants) | 2 | 9
  Dyspnoea: Week 81 | 11.11 (15.71) | -9.88 (22.53)
  Dyspnoea: Week 84: number analyzed (Participants) | 2 | 8
  Dyspnoea: Week 84 | 0.00 (0.00) | -6.94 (22.17)
  Dyspnoea: Week 87: number analyzed (Participants) | 1 | 4
  Dyspnoea: Week 87 | 0.00 | -2.78 (18.98)
  Dyspnoea: Week 90: number analyzed (Participants) | 1 | 2
  Dyspnoea: Week 90 | 0.00 | 5.56 (23.57)
  Dyspnoea: Week 93: number analyzed (Participants) | 0 | 1
  Dyspnoea: Week 93 |  | 22.22 (NA) — Only 1 participant.
  Dyspnoea: Time of First PD: number analyzed (Participants) | 61 | 70
  Dyspnoea: Time of First PD | 2.37 (22.05) | -0.16 (24.48)
  Dyspnoea: Time of Last Tx Dose: number analyzed (Participants) | 199 | 201
  Dyspnoea: Time of Last Tx Dose | 3.96 (22.74) | 0.44 (21.83)
  Dyspnoea: Survival Follow-Up Week 12: number analyzed (Participants) | 28 | 24
  Dyspnoea: Survival Follow-Up Week 12 | 9.92 (25.90) | 13.43 (33.73)
  Dyspnoea: Survival Follow-Up Week 24: number analyzed (Participants) | 19 | 7
  Dyspnoea: Survival Follow-Up Week 24 | 4.68 (17.50) | 4.76 (23.00)
  Pain In Chest: Week 3: number analyzed (Participants) | 213 | 205
  Pain In Chest: Week 3 | -1.25 (21.19) | 0.81 (23.67)
  Pain In Chest: Week 6: number analyzed (Participants) | 187 | 190
  Pain In Chest: Week 6 | 0.71 (25.15) | -6.32 (24.39)
  Pain In Chest: Week 9: number analyzed (Participants) | 162 | 173
  Pain In Chest: Week 9 | 0.82 (24.63) | -4.24 (25.57)
  Pain In Chest: Week 12: number analyzed (Participants) | 145 | 168
  Pain In Chest: Week 12 | -2.07 (24.60) | -0.60 (27.65)
  Pain In Chest: Week 15: number analyzed (Participants) | 137 | 159
  Pain In Chest: Week 15 | -1.46 (24.88) | -3.56 (25.60)
  Pain In Chest: Week 18: number analyzed (Participants) | 125 | 149
  Pain In Chest: Week 18 | -3.47 (26.38) | -3.36 (26.77)
  Pain In Chest: Week 21: number analyzed (Participants) | 100 | 146
  Pain In Chest: Week 21 | -3.33 (26.17) | -2.74 (25.22)
  Pain In Chest: Week 24: number analyzed (Participants) | 97 | 133
  Pain In Chest: Week 24 | -2.41 (26.89) | -4.76 (29.05)
  Pain In Chest: Week 27: number analyzed (Participants) | 78 | 123
  Pain In Chest: Week 27 | -5.13 (29.95) | -2.71 (22.82)
  Pain In Chest: Week 30: number analyzed (Participants) | 80 | 120
  Pain In Chest: Week 30 | -4.17 (29.71) | -3.06 (27.33)
  Pain In Chest: Week 33: number analyzed (Participants) | 72 | 103
  Pain In Chest: Week 33 | -0.46 (29.86) | -3.88 (28.12)
  Pain In Chest: Week 36: number analyzed (Participants) | 60 | 103
  Pain In Chest: Week 36 | -1.67 (31.55) | -2.91 (27.26)
  Pain In Chest: Week 39: number analyzed (Participants) | 60 | 92
  Pain In Chest: Week 39 | -3.89 (30.12) | -3.99 (27.44)
  Pain In Chest: Week 42: number analyzed (Participants) | 52 | 93
  Pain In Chest: Week 42 | -7.69 (29.24) | -7.17 (26.40)
  Pain In Chest: Week 45: number analyzed (Participants) | 48 | 77
  Pain In Chest: Week 45 | -6.25 (29.70) | -5.63 (25.02)
  Pain In Chest: Week 48: number analyzed (Participants) | 39 | 79
  Pain In Chest: Week 48 | -7.69 (29.08) | -4.64 (24.88)
  Pain In Chest: Week 51: number analyzed (Participants) | 36 | 79
  Pain In Chest: Week 51 | -11.11 (28.73) | -5.49 (24.13)
  Pain In Chest: Week 54: number analyzed (Participants) | 31 | 70
  Pain In Chest: Week 54 | -7.53 (29.45) | -4.29 (25.33)
  Pain In Chest: Week 57: number analyzed (Participants) | 26 | 69
  Pain In Chest: Week 57 | -1.28 (31.95) | -5.80 (26.17)
  Pain In Chest: Week 60: number analyzed (Participants) | 19 | 56
  Pain In Chest: Week 60 | 0.00 (22.22) | -3.57 (27.47)
  Pain In Chest: Week 63: number analyzed (Participants) | 13 | 39
  Pain In Chest: Week 63 | -5.13 (18.49) | -6.84 (25.57)
  Pain In Chest: Week 66: number analyzed (Participants) | 7 | 37
  Pain In Chest: Week 66 | -4.76 (23.00) | -4.50 (27.40)
  Pain In Chest: Week 69: number analyzed (Participants) | 6 | 28
  Pain In Chest: Week 69 | -16.67 (18.26) | -5.95 (31.50)
  Pain In Chest: Week 72: number analyzed (Participants) | 8 | 22
  Pain In Chest: Week 72 | -8.33 (23.57) | -4.55 (23.67)
  Pain In Chest: Week 75: number analyzed (Participants) | 5 | 23
  Pain In Chest: Week 75 | -6.67 (14.91) | 0.00 (20.10)
  Pain In Chest: Week 78: number analyzed (Participants) | 2 | 14
  Pain In Chest: Week 78 | 0.00 (0.00) | 0.00 (26.15)
  Pain In Chest: Week 81: number analyzed (Participants) | 2 | 9
  Pain In Chest: Week 81 | 0.00 (47.14) | 7.41 (14.70)
  Pain In Chest: Week 84: number analyzed (Participants) | 2 | 8
  Pain In Chest: Week 84 | 0.00 (0.00) | 4.17 (21.36)
  Pain In Chest: Week 87: number analyzed (Participants) | 1 | 4
  Pain In Chest: Week 87 | -33.33 (NA) — Only 1 participant. | 8.33 (16.67)
  Pain In Chest: Week 90: number analyzed (Participants) | 1 | 2
  Pain In Chest: Week 90 | -33.33 (NA) — Only 1 participant. | 0.00 (0.00)
  Pain In Chest: Week 93: number analyzed (Participants) | 0 | 1
  Pain In Chest: Week 93 |  | 0.00
  Pain In Chest: Time of First Pd: number analyzed (Participants) | 61 | 70
  Pain In Chest: Time of First Pd | 6.56 (22.62) | -3.81 (29.24)
  Pain In Chest: Time of Last Tx Dose: number analyzed (Participants) | 199 | 201
  Pain In Chest: Time of Last Tx Dose | 1.34 (25.26) | -0.83 (26.96)
  Pain In Chest: Survival Follow-Up Week 12: number analyzed (Participants) | 28 | 24
  Pain In Chest: Survival Follow-Up Week 12 | 5.95 (36.35) | -2.78 (32.48)
  Pain In Chest: Survival Follow-Up Week 24: number analyzed (Participants) | 19 | 7
  Pain In Chest: Survival Follow-Up Week 24 | 1.75 (17.48) | -4.76 (29.99)
  Pain In Arm Or Shoulder: Week 3: number analyzed (Participants) | 213 | 205
  Pain In Arm Or Shoulder: Week 3 | -4.69 (25.26) | -2.60 (24.78)
  Pain In Arm Or Shoulder: Week 6: number analyzed (Participants) | 187 | 190
  Pain In Arm Or Shoulder: Week 6 | -4.46 (23.14) | -5.44 (25.19)
  Pain In Arm Or Shoulder: Week 9: number analyzed (Participants) | 162 | 173
  Pain In Arm Or Shoulder: Week 9 | -2.88 (25.85) | -8.09 (28.73)
  Pain In Arm Or Shoulder: Week 12: number analyzed (Participants) | 145 | 168
  Pain In Arm Or Shoulder: Week 12 | -6.90 (23.54) | -4.37 (27.19)
  Pain In Arm Or Shoulder: Week 15: number analyzed (Participants) | 137 | 159
  Pain In Arm Or Shoulder: Week 15 | -3.89 (23.24) | -7.34 (30.15)
  Pain In Arm Or Shoulder: Week 18: number analyzed (Participants) | 125 | 149
  Pain In Arm Or Shoulder: Week 18 | -5.07 (25.77) | -6.26 (29.09)
  Pain In Arm Or Shoulder: Week 21: number analyzed (Participants) | 100 | 146
  Pain In Arm Or Shoulder: Week 21 | -6.00 (21.91) | -1.83 (28.71)
  Pain In Arm Or Shoulder: Week 24: number analyzed (Participants) | 97 | 133
  Pain In Arm Or Shoulder: Week 24 | -2.41 (28.16) | -5.26 (30.11)
  Pain In Arm Or Shoulder: Week 27: number analyzed (Participants) | 78 | 123
  Pain In Arm Or Shoulder: Week 27 | -5.56 (28.13) | -3.79 (26.72)
  Pain In Arm Or Shoulder: Week 30: number analyzed (Participants) | 80 | 120
  Pain In Arm Or Shoulder: Week 30 | 1.25 (27.27) | -3.33 (29.12)
  Pain In Arm Or Shoulder: Week 33: number analyzed (Participants) | 72 | 103
  Pain In Arm Or Shoulder: Week 33 | -5.56 (25.02) | -1.94 (27.54)
  Pain In Arm Or Shoulder: Week 36: number analyzed (Participants) | 60 | 103
  Pain In Arm Or Shoulder: Week 36 | -1.67 (30.33) | -3.24 (31.49)
  Pain In Arm Or Shoulder: Week 39: number analyzed (Participants) | 60 | 92
  Pain In Arm Or Shoulder: Week 39 | -5.00 (30.58) | -3.99 (30.80)
  Pain In Arm Or Shoulder: Week 42: number analyzed (Participants) | 52 | 93
  Pain In Arm Or Shoulder: Week 42 | 0.00 (28.77) | -8.60 (25.49)
  Pain In Arm Or Shoulder: Week 45: number analyzed (Participants) | 48 | 77
  Pain In Arm Or Shoulder: Week 45 | -0.69 (27.06) | -6.06 (28.47)
  Pain In Arm Or Shoulder: Week 48: number analyzed (Participants) | 39 | 79
  Pain In Arm Or Shoulder: Week 48 | -1.71 (27.52) | -4.22 (29.89)
  Pain In Arm Or Shoulder: Week 51: number analyzed (Participants) | 36 | 79
  Pain In Arm Or Shoulder: Week 51 | -2.78 (25.67) | -3.38 (27.53)
  Pain In Arm Or Shoulder: Week 54: number analyzed (Participants) | 31 | 70
  Pain In Arm Or Shoulder: Week 54 | -1.08 (21.92) | -6.19 (25.56)
  Pain In Arm Or Shoulder: Week 57: number analyzed (Participants) | 26 | 69
  Pain In Arm Or Shoulder: Week 57 | -1.28 (22.07) | -2.90 (26.65)
  Pain In Arm Or Shoulder: Week 60: number analyzed (Participants) | 19 | 56
  Pain In Arm Or Shoulder: Week 60 | -5.26 (20.07) | -4.17 (27.75)
  Pain In Arm Or Shoulder: Week 63: number analyzed (Participants) | 13 | 39
  Pain In Arm Or Shoulder: Week 63 | -5.13 (18.49) | -3.42 (27.35)
  Pain In Arm Or Shoulder: Week 66: number analyzed (Participants) | 7 | 37
  Pain In Arm Or Shoulder: Week 66 | 4.76 (12.60) | -1.80 (31.37)
  Pain In Arm Or Shoulder: Week 69: number analyzed (Participants) | 6 | 28
  Pain In Arm Or Shoulder: Week 69 | 0.00 (0.00) | -7.14 (22.87)
  Pain In Arm Or Shoulder: Week 72: number analyzed (Participants) | 8 | 22
  Pain In Arm Or Shoulder: Week 72 | -8.33 (15.43) | -7.58 (27.08)
  Pain In Arm Or Shoulder: Week 75: number analyzed (Participants) | 5 | 23
  Pain In Arm Or Shoulder: Week 75 | -6.67 (14.91) | -8.70 (25.06)
  Pain In Arm Or Shoulder: Week 78: number analyzed (Participants) | 2 | 14
  Pain In Arm Or Shoulder: Week 78 | 0.00 (0.00) | -2.38 (24.33)
  Pain In Arm Or Shoulder: Week 81: number analyzed (Participants) | 2 | 9
  Pain In Arm Or Shoulder: Week 81 | 0.00 (0.00) | 3.70 (11.11)
  Pain In Arm Or Shoulder: Week 84: number analyzed (Participants) | 2 | 8
  Pain In Arm Or Shoulder: Week 84 | 0.00 (0.00) | 4.17 (21.36)
  Pain In Arm Or Shoulder: Week 87: number analyzed (Participants) | 1 | 4
  Pain In Arm Or Shoulder: Week 87 | 0.00 (NA) — Only 1 participant. | -16.67 (33.33)
  Pain In Arm Or Shoulder: Week 90: number analyzed (Participants) | 1 | 2
  Pain In Arm Or Shoulder: Week 90 | 0.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Pain In Arm Or Shoulder: Week 93: number analyzed (Participants) | 0 | 1
  Pain In Arm Or Shoulder: Week 93 |  | 0.00 (NA) — Only 1 participant.
  Pain In Arm Or Shoulder: Time of First Pd: number analyzed (Participants) | 61 | 70
  Pain In Arm Or Shoulder: Time of First Pd | 2.19 (28.46) | 1.90 (25.94)
  Pain In Arm Or Shoulder: Time of Last Tx Dose: number analyzed (Participants) | 199 | 201
  Pain In Arm Or Shoulder: Time of Last Tx Dose | -0.50 (27.11) | 0.33 (30.55)
  Pain In Arm Or Shoulder:Survival Follow-Up Week 12: number analyzed (Participants) | 28 | 24
  Pain In Arm Or Shoulder:Survival Follow-Up Week 12 | 13.10 (30.55) | 5.56 (40.13)
  Pain In Arm Or Shoulder:Survival Follow-Up Week 24: number analyzed (Participants) | 19 | 7
  Pain In Arm Or Shoulder:Survival Follow-Up Week 24 | 1.75 (28.27) | 0.00 (0.00)

9. Secondary Outcome: Change From Baseline in Patient-Reported Lung Cancer Symptoms as Reported Using the Symptoms in Lung Cancer (SILC) Scale Score
Description: Change from baseline per SILC scale will be analyzed for each lung cancer symptoms scores. SILC questionnaire comprises 3 individual symptoms & are scored at individual symptom level, thus have a dyspnea score, chest pain score, & cough score. There are a total of 9 questions in SILC questionnaire, each question has a minimum value of 0 & maximum value of 4. Each individual symptom score is calculated as average of responses for symptom items. 'Chest pain' score is mean of question 1 & 2, 'Cough' score is mean of question 3 & 4 and 'Dyspnea' score is mean of question 5 to 9 in SILC questionnaire. An increase in score is suggestive of a worsening in symptomology. A score change of ≥0.3 points for dyspnea & cough symptom scores is considered to be clinically significant; whereas a score change of≥0.5 points for chest pain score is considered to be clinically significant.
Time Frame: Baseline up to 3 and 6 months after disease progression or loss of clinical benefit (up to approximately 25 months)
Population: ITT population with a non-missing baseline and at least a post-baseline PRO assessment (i.e., PRO evaluable population).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 176 | 200
Units on a scale
  Chest Pain: Week 1: number analyzed (Participants) | 160 | 186
  Chest Pain: Week 1 | 0.20 (0.83) | 0.30 (0.88)
  Chest Pain: Week 2: number analyzed (Participants) | 152 | 176
  Chest Pain: Week 2 | -0.01 (0.88) | 0.21 (0.85)
  Chest Pain: Week 3: number analyzed (Participants) | 151 | 165
  Chest Pain: Week 3 | -0.05 (0.92) | 0.06 (0.95)
  Chest Pain: Week 4: number analyzed (Participants) | 144 | 160
  Chest Pain: Week 4 | 0.03 (0.91) | 0.03 (0.93)
  Chest Pain: Week 5: number analyzed (Participants) | 143 | 166
  Chest Pain: Week 5 | -0.02 (0.93) | -0.01 (0.88)
  Chest Pain: Week 6: number analyzed (Participants) | 132 | 166
  Chest Pain: Week 6 | -0.05 (0.88) | -0.02 (0.92)
  Chest Pain: Week 7: number analyzed (Participants) | 132 | 156
  Chest Pain: Week 7 | 0.07 (1.00) | -0.04 (1.00)
  Chest Pain: Week 8: number analyzed (Participants) | 124 | 157
  Chest Pain: Week 8 | 0.03 (0.94) | -0.07 (1.02)
  Chest Pain: Week 9: number analyzed (Participants) | 125 | 159
  Chest Pain: Week 9 | 0.06 (1.00) | -0.03 (1.03)
  Chest Pain: Week 10: number analyzed (Participants) | 120 | 152
  Chest Pain: Week 10 | 0.03 (1.02) | 0.02 (1.05)
  Chest Pain: Week 11: number analyzed (Participants) | 117 | 156
  Chest Pain: Week 11 | 0.02 (0.96) | 0.04 (1.09)
  Chest Pain: Week 12: number analyzed (Participants) | 116 | 142
  Chest Pain: Week 12 | -0.02 (0.96) | -0.01 (1.02)
  Chest Pain: Week 13: number analyzed (Participants) | 108 | 142
  Chest Pain: Week 13 | -0.05 (1.02) | 0.05 (0.97)
  Chest Pain: Week 14: number analyzed (Participants) | 103 | 132
  Chest Pain: Week 14 | -0.07 (1.12) | 0.06 (1.06)
  Chest Pain: Week 15: number analyzed (Participants) | 101 | 133
  Chest Pain: Week 15 | 0.13 (1.16) | 0.08 (0.94)
  Chest Pain: Week 16: number analyzed (Participants) | 100 | 133
  Chest Pain: Week 16 | 0.02 (1.08) | 0.08 (1.04)
  Chest Pain: Week 17: number analyzed (Participants) | 97 | 131
  Chest Pain: Week 17 | 0.02 (1.08) | 0.00 (1.08)
  Chest Pain: Week 18: number analyzed (Participants) | 88 | 121
  Chest Pain: Week 18 | -0.06 (1.11) | 0.12 (1.07)
  Chest Pain: Week 19: number analyzed (Participants) | 81 | 122
  Chest Pain: Week 19 | -0.15 (1.12) | 0.02 (1.01)
  Chest Pain: Week 20: number analyzed (Participants) | 71 | 112
  Chest Pain: Week 20 | -0.02 (1.22) | -0.01 (1.03)
  Chest Pain: Week 21: number analyzed (Participants) | 74 | 114
  Chest Pain: Week 21 | 0.03 (1.28) | 0.01 (1.03)
  Chest Pain: Week 22: number analyzed (Participants) | 65 | 106
  Chest Pain: Week 22 | 0.04 (1.21) | 0.02 (1.02)
  Chest Pain: Week 23: number analyzed (Participants) | 65 | 106
  Chest Pain: Week 23 | -0.08 (1.14) | 0.04 (0.96)
  Chest Pain: Week 24: number analyzed (Participants) | 64 | 106
  Chest Pain: Week 24 | -0.02 (1.16) | 0.09 (0.99)
  Chest Pain: Week 25: number analyzed (Participants) | 60 | 100
  Chest Pain: Week 25 | 0.05 (1.24) | 0.14 (1.03)
  Chest Pain: Week 26: number analyzed (Participants) | 55 | 100
  Chest Pain: Week 26 | -0.05 (1.14) | 0.09 (1.00)
  Chest Pain: Week 27: number analyzed (Participants) | 55 | 99
  Chest Pain: Week 27 | 0.04 (1.17) | 0.04 (1.01)
  Chest Pain: Week 28: number analyzed (Participants) | 55 | 96
  Chest Pain: Week 28 | 0.24 (1.18) | 0.03 (0.93)
  Chest Pain: Week 29: number analyzed (Participants) | 54 | 99
  Chest Pain: Week 29 | 0.06 (1.29) | 0.04 (0.95)
  Chest Pain: Week 30: number analyzed (Participants) | 52 | 95
  Chest Pain: Week 30 | 0.01 (1.37) | 0.04 (0.97)
  Chest Pain: Week 31: number analyzed (Participants) | 44 | 93
  Chest Pain: Week 31 | 0.02 (1.09) | 0.05 (0.88)
  Chest Pain: Week 32: number analyzed (Participants) | 39 | 94
  Chest Pain: Week 32 | 0.21 (1.21) | -0.01 (0.98)
  Chest Pain: Week 33: number analyzed (Participants) | 41 | 85
  Chest Pain: Week 33 | 0.04 (1.17) | 0.03 (0.92)
  Chest Pain: Week 34: number analyzed (Participants) | 40 | 84
  Chest Pain: Week 34 | 0.21 (1.27) | 0.11 (0.99)
  Chest Pain: Week 35: number analyzed (Participants) | 39 | 87
  Chest Pain: Week 35 | 0.33 (1.30) | 0.11 (0.98)
  Chest Pain: Week 36: number analyzed (Participants) | 34 | 86
  Chest Pain: Week 36 | 0.15 (1.07) | 0.17 (1.04)
  Chest Pain: Week 37: number analyzed (Participants) | 33 | 86
  Chest Pain: Week 37 | 0.15 (1.21) | 0.06 (0.94)
  Chest Pain: Week 38: number analyzed (Participants) | 30 | 80
  Chest Pain: Week 38 | 0.12 (1.16) | 0.04 (1.03)
  Chest Pain: Week 39: number analyzed (Participants) | 32 | 72
  Chest Pain: Week 39 | 0.20 (1.23) | 0.13 (1.01)
  Chest Pain: Week 40: number analyzed (Participants) | 31 | 77
  Chest Pain: Week 40 | 0.15 (1.31) | 0.04 (0.96)
  Chest Pain: Week 41: number analyzed (Participants) | 30 | 74
  Chest Pain: Week 41 | -0.05 (1.06) | 0.09 (1.03)
  Chest Pain: Week 42: number analyzed (Participants) | 27 | 73
  Chest Pain: Week 42 | -0.06 (1.07) | 0.03 (1.02)
  Chest Pain: Week 43: number analyzed (Participants) | 23 | 76
  Chest Pain: Week 43 | -0.22 (0.82) | 0.13 (1.02)
  Chest Pain: Week 44: number analyzed (Participants) | 25 | 72
  Chest Pain: Week 44 | -0.10 (1.29) | 0.10 (1.04)
  Chest Pain: Week 45: number analyzed (Participants) | 25 | 69
  Chest Pain: Week 45 | -0.20 (1.24) | 0.03 (0.95)
  Chest Pain: Week 46: number analyzed (Participants) | 24 | 67
  Chest Pain: Week 46 | -0.06 (1.18) | 0.08 (0.99)
  Chest Pain: Week 47: number analyzed (Participants) | 23 | 63
  Chest Pain: Week 47 | 0.02 (1.09) | 0.09 (0.91)
  Chest Pain: Week 48: number analyzed (Participants) | 25 | 64
  Chest Pain: Week 48 | 0.02 (1.27) | 0.05 (1.00)
  Chest Pain: Week 49: number analyzed (Participants) | 23 | 62
  Chest Pain: Week 49 | -0.09 (1.07) | 0.03 (0.90)
  Chest Pain: Week 50: number analyzed (Participants) | 23 | 58
  Chest Pain: Week 50 | -0.13 (0.99) | 0.00 (1.03)
  Chest Pain: Week 51: number analyzed (Participants) | 21 | 62
  Chest Pain: Week 51 | -0.02 (0.77) | 0.12 (0.94)
  Chest Pain: Week 52: number analyzed (Participants) | 21 | 55
  Chest Pain: Week 52 | 0.14 (1.06) | 0.00 (1.11)
  Chest Pain: Week 53: number analyzed (Participants) | 23 | 54
  Chest Pain: Week 53 | 0.13 (1.35) | -0.01 (1.06)
  Chest Pain: Week 54: number analyzed (Participants) | 22 | 54
  Chest Pain: Week 54 | 0.11 (1.16) | -0.08 (1.10)
  Chest Pain: Week 55: number analyzed (Participants) | 21 | 49
  Chest Pain: Week 55 | 0.12 (1.38) | 0.03 (1.14)
  Chest Pain: Week 56: number analyzed (Participants) | 20 | 53
  Chest Pain: Week 56 | 0.13 (1.46) | 0.04 (1.18)
  Chest Pain: Week 57: number analyzed (Participants) | 17 | 46
  Chest Pain: Week 57 | 0.12 (1.21) | -0.01 (1.15)
  Chest Pain: Week 58: number analyzed (Participants) | 15 | 43
  Chest Pain: Week 58 | 0.27 (0.98) | -0.12 (1.10)
  Chest Pain: Week 59: number analyzed (Participants) | 13 | 40
  Chest Pain: Week 59 | 0.23 (0.73) | -0.23 (1.01)
  Chest Pain: Week 60: number analyzed (Participants) | 11 | 41
  Chest Pain: Week 60 | 0.14 (0.67) | -0.15 (1.17)
  Chest Pain: Week 61: number analyzed (Participants) | 13 | 43
  Chest Pain: Week 61 | 0.23 (0.83) | 0.00 (1.06)
  Chest Pain: Week 62: number analyzed (Participants) | 13 | 37
  Chest Pain: Week 62 | 0.46 (0.72) | -0.04 (1.08)
  Chest Pain: Week 63: number analyzed (Participants) | 12 | 36
  Chest Pain: Week 63 | 0.25 (0.75) | -0.06 (1.09)
  Chest Pain: Week 64: number analyzed (Participants) | 10 | 35
  Chest Pain: Week 64 | 0.15 (0.78) | 0.09 (0.95)
  Chest Pain: Week 65: number analyzed (Participants) | 9 | 33
  Chest Pain: Week 65 | 0.11 (0.82) | -0.03 (0.99)
  Chest Pain: Week 66: number analyzed (Participants) | 6 | 34
  Chest Pain: Week 66 | 0.42 (0.92) | 0.13 (1.05)
  Chest Pain: Week 67: number analyzed (Participants) | 7 | 30
  Chest Pain: Week 67 | 0.36 (0.85) | 0.02 (1.00)
  Chest Pain: Week 68: number analyzed (Participants) | 6 | 30
  Chest Pain: Week 68 | 0.33 (0.88) | 0.12 (1.18)
  Chest Pain: Week 69: number analyzed (Participants) | 7 | 29
  Chest Pain: Week 69 | 0.07 (0.93) | -0.05 (1.10)
  Chest Pain: Week 70: number analyzed (Participants) | 6 | 30
  Chest Pain: Week 70 | 0.25 (0.88) | 0.03 (1.11)
  Chest Pain: Week 71: number analyzed (Participants) | 5 | 26
  Chest Pain: Week 71 | 0.30 (0.97) | 0.04 (1.09)
  Chest Pain: Week 72: number analyzed (Participants) | 4 | 25
  Chest Pain: Week 72 | -0.13 (0.25) | -0.22 (0.94)
  Chest Pain: Week 73: number analyzed (Participants) | 4 | 24
  Chest Pain: Week 73 | 0.13 (1.31) | -0.10 (1.01)
  Chest Pain: Week 74: number analyzed (Participants) | 4 | 23
  Chest Pain: Week 74 | 0.38 (1.11) | -0.02 (1.14)
  Chest Pain: Week 75: number analyzed (Participants) | 4 | 21
  Chest Pain: Week 75 | 0.38 (1.11) | -0.07 (1.14)
  Chest Pain: Week 76: number analyzed (Participants) | 3 | 17
  Chest Pain: Week 76 | 0.00 (0.50) | -0.06 (1.20)
  Chest Pain: Week 77: number analyzed (Participants) | 2 | 17
  Chest Pain: Week 77 | -0.25 (0.35) | -0.21 (1.03)
  Chest Pain: Week 78: number analyzed (Participants) | 2 | 14
  Chest Pain: Week 78 | -0.75 (0.35) | -0.25 (1.14)
  Chest Pain: Week 79: number analyzed (Participants) | 2 | 14
  Chest Pain: Week 79 | 0.00 (0.71) | -0.18 (1.20)
  Chest Pain: Week 80: number analyzed (Participants) | 2 | 13
  Chest Pain: Week 80 | -0.25 (0.35) | -0.12 (0.96)
  Chest Pain: Week 81: number analyzed (Participants) | 2 | 12
  Chest Pain: Week 81 | -0.25 (0.35) | -0.25 (0.89)
  Chest Pain: Week 82: number analyzed (Participants) | 2 | 9
  Chest Pain: Week 82 | -0.75 (0.35) | 0.00 (1.25)
  Chest Pain: Week 83: number analyzed (Participants) | 2 | 4
  Chest Pain: Week 83 | -0.25 (0.35) | -0.50 (1.73)
  Chest Pain: Week 84: number analyzed (Participants) | 2 | 5
  Chest Pain: Week 84 | 0.00 (0.71) | -0.30 (1.57)
  Chest Pain: Week 85: number analyzed (Participants) | 1 | 5
  Chest Pain: Week 85 | -1.00 (NA) — Only 1 participant. | -0.20 (1.68)
  Chest Pain: Week 86: number analyzed (Participants) | 1 | 4
  Chest Pain: Week 86 | 0.00 (NA) — Only 1 participant. | -0.50 (1.73)
  Chest Pain: Week 87: number analyzed (Participants) | 1 | 3
  Chest Pain: Week 87 | -1.00 (NA) — Only 1 participant. | 0.50 (0.87)
  Chest Pain: Week 88: number analyzed (Participants) | 1 | 4
  Chest Pain: Week 88 | -1.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Chest Pain: Week 89: number analyzed (Participants) | 1 | 2
  Chest Pain: Week 89 | -1.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Chest Pain: Week 90: number analyzed (Participants) | 1 | 2
  Chest Pain: Week 90 | 0.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Chest Pain: Week 91: number analyzed (Participants) | 1 | 2
  Chest Pain: Week 91 | 0.00 (NA) — Only 1 participant. | 0.00 (0.00)
  Chest Pain: Week 92: number analyzed (Participants) | 0 | 2
  Chest Pain: Week 92 |  | 0.00 (0.00)
  Chest Pain: Week 93: number analyzed (Participants) | 0 | 2
  Chest Pain: Week 93 |  | 0.00 (0.00)
  Chest Pain: Week 94: number analyzed (Participants) | 0 | 1
  Chest Pain: Week 94 |  | 1.00 (NA) — Only 1 participant.
  Chest Pain: Week 95: number analyzed (Participants) | 0 | 1
  Chest Pain: Week 95 |  | 0.50 (NA) — Only 1 participant.
  Chest Pain: Time of First Pd: number analyzed (Participants) | 110 | 96
  Chest Pain: Time of First Pd | 0.28 (1.06) | 0.20 (0.91)
  Chest Pain: Time of Last Tx Dose: number analyzed (Participants) | 141 | 150
  Chest Pain: Time of Last Tx Dose | 0.17 (1.17) | 0.13 (0.98)
  Cough: Week 1: number analyzed (Participants) | 160 | 186
  Cough: Week 1 | -0.08 (0.74) | -0.06 (0.89)
  Cough: Week 2: number analyzed (Participants) | 152 | 176
  Cough: Week 2 | -0.13 (0.73) | -0.08 (0.90)
  Cough: Week 3: number analyzed (Participants) | 151 | 165
  Cough: Week 3 | -0.05 (0.77) | -0.07 (0.81)
  Cough: Week 4: number analyzed (Participants) | 144 | 160
  Cough: Week 4 | -0.11 (0.89) | -0.22 (0.85)
  Cough: Week 5: number analyzed (Participants) | 143 | 166
  Cough: Week 5 | -0.14 (0.83) | -0.33 (0.89)
  Cough: Week 6: number analyzed (Participants) | 132 | 166
  Cough: Week 6 | -0.16 (0.85) | -0.33 (0.91)
  Cough: Week 7: number analyzed (Participants) | 132 | 156
  Cough: Week 7 | -0.22 (0.89) | -0.22 (0.97)
  Cough: Week 8: number analyzed (Participants) | 124 | 157
  Cough: Week 8 | -0.20 (0.89) | -0.28 (0.98)
  Cough: Week 9: number analyzed (Participants) | 125 | 159
  Cough: Week 9 | -0.17 (0.91) | -0.29 (0.97)
  Cough: Week 10: number analyzed (Participants) | 120 | 152
  Cough: Week 10 | -0.22 (0.95) | -0.35 (1.06)
  Cough: Week 11: number analyzed (Participants) | 117 | 156
  Cough: Week 11 | -0.21 (0.99) | -0.33 (1.02)
  Cough: Week 12: number analyzed (Participants) | 116 | 142
  Cough: Week 12 | -0.13 (1.05) | -0.40 (0.96)
  Cough: Week 13: number analyzed (Participants) | 108 | 142
  Cough: Week 13 | -0.24 (1.05) | -0.37 (1.04)
  Cough: Week 14: number analyzed (Participants) | 103 | 132
  Cough: Week 14 | -0.23 (0.98) | -0.34 (1.03)
  Cough: Week 15: number analyzed (Participants) | 101 | 133
  Cough: Week 15 | -0.11 (1.03) | -0.33 (1.03)
  Cough: Week 16: number analyzed (Participants) | 100 | 133
  Cough: Week 16 | -0.20 (1.05) | -0.33 (1.04)
  Cough: Week 17: number analyzed (Participants) | 97 | 131
  Cough: Week 17 | -0.20 (1.11) | -0.31 (0.99)
  Cough: Week 18: number analyzed (Participants) | 88 | 121
  Cough: Week 18 | -0.19 (1.12) | -0.31 (1.00)
  Cough: Week 19: number analyzed (Participants) | 81 | 122
  Cough: Week 19 | -0.25 (1.07) | -0.36 (1.06)
  Cough: Week 20: number analyzed (Participants) | 71 | 112
  Cough: Week 20 | -0.25 (1.16) | -0.39 (0.99)
  Cough: Week 21: number analyzed (Participants) | 74 | 114
  Cough: Week 21 | -0.19 (1.09) | -0.36 (1.07)
  Cough: Week 22: number analyzed (Participants) | 65 | 106
  Cough: Week 22 | -0.29 (1.11) | -0.41 (1.08)
  Cough: Week 23: number analyzed (Participants) | 65 | 106
  Cough: Week 23 | -0.34 (1.07) | -0.44 (1.04)
  Cough: Week 24: number analyzed (Participants) | 64 | 106
  Cough: Week 24 | -0.27 (0.96) | -0.29 (1.13)
  Cough: Week 25: number analyzed (Participants) | 60 | 100
  Cough: Week 25 | -0.24 (1.11) | -0.27 (1.10)
  Cough: Week 26: number analyzed (Participants) | 55 | 100
  Cough: Week 26 | -0.25 (1.16) | -0.22 (1.22)
  Cough: Week 27: number analyzed (Participants) | 55 | 99
  Cough: Week 27 | -0.19 (0.99) | -0.32 (1.11)
  Cough: Week 28: number analyzed (Participants) | 55 | 96
  Cough: Week 28 | -0.19 (1.04) | -0.32 (1.12)
  Cough: Week 29: number analyzed (Participants) | 54 | 99
  Cough: Week 29 | -0.25 (1.13) | -0.34 (1.11)
  Cough: Week 30: number analyzed (Participants) | 52 | 95
  Cough: Week 30 | -0.08 (1.12) | -0.34 (1.00)
  Cough: Week 31: number analyzed (Participants) | 44 | 93
  Cough: Week 31 | -0.13 (1.13) | -0.37 (0.99)
  Cough: Week 32: number analyzed (Participants) | 39 | 94
  Cough: Week 32 | 0.01 (1.09) | -0.45 (0.94)
  Cough: Week 33: number analyzed (Participants) | 41 | 85
  Cough: Week 33 | 0.05 (1.17) | -0.44 (0.99)
  Cough: Week 34: number analyzed (Participants) | 40 | 84
  Cough: Week 34 | -0.10 (1.09) | -0.29 (1.02)
  Cough: Week 35: number analyzed (Participants) | 39 | 87
  Cough: Week 35 | -0.27 (1.05) | -0.32 (0.99)
  Cough: Week 36: number analyzed (Participants) | 34 | 86
  Cough: Week 36 | 0.01 (1.10) | -0.31 (0.99)
  Cough: Week 37: number analyzed (Participants) | 33 | 86
  Cough: Week 37 | -0.11 (1.16) | -0.37 (1.01)
  Cough: Week 38: number analyzed (Participants) | 30 | 80
  Cough: Week 38 | 0.02 (1.03) | -0.31 (1.03)
  Cough: Week 39: number analyzed (Participants) | 32 | 72
  Cough: Week 39 | 0.02 (1.19) | -0.33 (0.98)
  Cough: Week 40: number analyzed (Participants) | 31 | 77
  Cough: Week 40 | -0.10 (1.15) | -0.35 (1.07)
  Cough: Week 41: number analyzed (Participants) | 30 | 74
  Cough: Week 41 | -0.27 (1.10) | -0.30 (1.09)
  Cough: Week 42: number analyzed (Participants) | 27 | 73
  Cough: Week 42 | -0.31 (1.04) | -0.31 (1.04)
  Cough: Week 43: number analyzed (Participants) | 23 | 76
  Cough: Week 43 | -0.20 (1.04) | -0.37 (0.98)
  Cough: Week 44: number analyzed (Participants) | 25 | 72
  Cough: Week 44 | 0.00 (1.04) | -0.36 (1.03)
  Cough: Week 45: number analyzed (Participants) | 25 | 69
  Cough: Week 45 | -0.18 (1.14) | -0.41 (1.04)
  Cough: Week 46: number analyzed (Participants) | 24 | 67
  Cough: Week 46 | -0.25 (1.04) | -0.34 (1.17)
  Cough: Week 47: number analyzed (Participants) | 23 | 63
  Cough: Week 47 | -0.43 (1.09) | -0.29 (1.17)
  Cough: Week 48: number analyzed (Participants) | 25 | 64
  Cough: Week 48 | -0.26 (1.16) | -0.38 (1.08)
  Cough: Week 49: number analyzed (Participants) | 23 | 62
  Cough: Week 49 | -0.50 (1.07) | -0.40 (1.10)
  Cough: Week 50: number analyzed (Participants) | 23 | 58
  Cough: Week 50 | -0.37 (0.84) | -0.40 (1.06)
  Cough: Week 51: number analyzed (Participants) | 21 | 62
  Cough: Week 51 | -0.45 (1.16) | -0.15 (1.10)
  Cough: Week 52: number analyzed (Participants) | 21 | 55
  Cough: Week 52 | -0.29 (1.07) | -0.10 (1.17)
  Cough: Week 53: number analyzed (Participants) | 23 | 54
  Cough: Week 53 | -0.24 (1.21) | -0.13 (1.17)
  Cough: Week 54: number analyzed (Participants) | 22 | 54
  Cough: Week 54 | -0.27 (1.10) | -0.16 (1.15)
  Cough: Week 55: number analyzed (Participants) | 21 | 49
  Cough: Week 55 | -0.10 (1.15) | -0.35 (1.13)
  Cough: Week 56: number analyzed (Participants) | 20 | 53
  Cough: Week 56 | -0.30 (1.14) | -0.26 (1.17)
  Cough: Week 57: number analyzed (Participants) | 17 | 46
  Cough: Week 57 | -0.41 (0.92) | -0.25 (1.10)
  Cough: Week 58: number analyzed (Participants) | 15 | 43
  Cough: Week 58 | -0.17 (1.05) | -0.45 (0.96)
  Cough: Week 59: number analyzed (Participants) | 13 | 40
  Cough: Week 59 | -0.31 (0.93) | -0.50 (1.02)
  Cough: Week 60: number analyzed (Participants) | 11 | 41
  Cough: Week 60 | -0.55 (1.04) | -0.52 (1.03)
  Cough: Week 61: number analyzed (Participants) | 13 | 43
  Cough: Week 61 | -0.23 (1.15) | -0.38 (1.07)
  Cough: Week 62: number analyzed (Participants) | 13 | 37
  Cough: Week 62 | 0.04 (1.03) | -0.53 (1.15)
  Cough: Week 63: number analyzed (Participants) | 12 | 36
  Cough: Week 63 | -0.29 (1.18) | -0.57 (1.10)
  Cough: Week 64: number analyzed (Participants) | 10 | 35
  Cough: Week 64 | -0.45 (1.04) | -0.49 (1.01)
  Cough: Week 65: number analyzed (Participants) | 9 | 33
  Cough: Week 65 | -0.61 (0.96) | -0.39 (0.94)
  Cough: Week 66: number analyzed (Participants) | 6 | 34
  Cough: Week 66 | -0.17 (0.82) | -0.43 (1.18)
  Cough: Week 67: number analyzed (Participants) | 7 | 30
  Cough: Week 67 | -0.64 (1.07) | -0.47 (0.84)
  Cough: Week 68: number analyzed (Participants) | 6 | 30
  Cough: Week 68 | -0.75 (0.88) | -0.35 (1.04)
  Cough: Week 69: number analyzed (Participants) | 7 | 29
  Cough: Week 69 | -0.57 (1.10) | -0.53 (0.90)
  Cough: Week 70: number analyzed (Participants) | 6 | 30
  Cough: Week 70 | -0.83 (0.93) | -0.43 (0.98)
  Cough: Week 71: number analyzed (Participants) | 5 | 26
  Cough: Week 71 | -0.90 (0.89) | -0.56 (1.04)
  Cough: Week 72: number analyzed (Participants) | 4 | 25
  Cough: Week 72 | -1.25 (0.50) | -0.72 (1.15)
  Cough: Week 73: number analyzed (Participants) | 4 | 24
  Cough: Week 73 | -0.63 (1.11) | -0.77 (1.00)
  Cough: Week 74: number analyzed (Participants) | 4 | 23
  Cough: Week 74 | -0.63 (1.11) | -0.54 (0.94)
  Cough: Week 75: number analyzed (Participants) | 4 | 21
  Cough: Week 75 | -0.63 (1.11) | -0.67 (1.00)
  Cough: Week 76: number analyzed (Participants) | 3 | 17
  Cough: Week 76 | -1.00 (1.00) | -0.65 (1.22)
  Cough: Week 77: number analyzed (Participants) | 2 | 17
  Cough: Week 77 | -0.50 (0.71) | -0.82 (1.21)
  Cough: Week 78: number analyzed (Participants) | 2 | 14
  Cough: Week 78 | -1.00 (0.00) | -0.57 (1.04)
  Cough: Week 79: number analyzed (Participants) | 2 | 14
  Cough: Week 79 | -0.25 (0.35) | -0.64 (1.23)
  Cough: Week 80: number analyzed (Participants) | 2 | 13
  Cough: Week 80 | -0.50 (0.71) | -1.04 (1.11)
  Cough: Week 81: number analyzed (Participants) | 2 | 12
  Cough: Week 81 | -0.50 (0.71) | -0.79 (1.05)
  Cough: Week 82: number analyzed (Participants) | 2 | 9
  Cough: Week 82 | -0.50 (0.71) | -0.89 (1.27)
  Cough: Week 83: number analyzed (Participants) | 2 | 4
  Cough: Week 83 | -1.00 (0.00) | 0.13 (1.03)
  Cough: Week 84: number analyzed (Participants) | 2 | 5
  Cough: Week 84 | -0.50 (0.71) | -0.20 (1.04)
  Cough: Week 85: number analyzed (Participants) | 1 | 5
  Cough: Week 85 | 0.00 (NA) — Only 1 participant. | 0.00 (0.87)
  Cough: Week 86: number analyzed (Participants) | 1 | 4
  Cough: Week 86 | 0.00 (NA) — Only 1 participant. | -0.38 (0.48)
  Cough: Week 87: number analyzed (Participants) | 1 | 3
  Cough: Week 87 | 0.00 (NA) — Only 1 participant. | -0.83 (0.58)
  Cough: Week 88: number analyzed (Participants) | 1 | 4
  Cough: Week 88 | 0.00 (NA) — Only 1 participant. | -0.88 (0.48)
  Cough: Week 89: number analyzed (Participants) | 1 | 2
  Cough: Week 89 | 0.00 | 0.00 (0.71)
  Cough: Week 90: number analyzed (Participants) | 1 | 2
  Cough: Week 90 | 0.00 | 0.25 (1.06)
  Cough: Week 91: number analyzed (Participants) | 1 | 2
  Cough: Week 91 | 0.00 | -0.50 (0.00)
  Cough: Week 92: number analyzed (Participants) | 0 | 2
  Cough: Week 92 |  | 0.50 (0.71)
  Cough: Week 93: number analyzed (Participants) | 0 | 2
  Cough: Week 93 |  | 0.50 (0.71)
  Cough: Week 94: number analyzed (Participants) | 0 | 1
  Cough: Week 94 |  | 0.50 (NA) — Only 1 participant.
  Cough: Week 95: number analyzed (Participants) | 0 | 1
  Cough: Week 95 |  | 0.00 (NA) — Only 1 participant.
  Cough: Time of First Pd: number analyzed (Participants) | 110 | 96
  Cough: Time of First Pd | -0.08 (1.12) | -0.45 (0.93)
  Cough: Time of Last Tx Dose: number analyzed (Participants) | 141 | 150
  Cough: Time of Last Tx Dose | -0.15 (0.95) | -0.29 (0.91)
  Dyspnoea: Week 1: number analyzed (Participants) | 160 | 186
  Dyspnoea: Week 1 | 0.20 (0.82) | 0.16 (0.81)
  Dyspnoea: Week 2: number analyzed (Participants) | 152 | 176
  Dyspnoea: Week 2 | 0.11 (0.76) | 0.15 (0.82)
  Dyspnoea: Week 3: number analyzed (Participants) | 151 | 165
  Dyspnoea: Week 3 | 0.10 (0.71) | 0.12 (0.70)
  Dyspnoea: Week 4: number analyzed (Participants) | 144 | 160
  Dyspnoea: Week 4 | 0.21 (0.84) | 0.17 (0.95)
  Dyspnoea: Week 5: number analyzed (Participants) | 143 | 166
  Dyspnoea: Week 5 | 0.22 (0.82) | 0.17 (0.91)
  Dyspnoea: Week 6: number analyzed (Participants) | 132 | 166
  Dyspnoea: Week 6 | 0.23 (0.82) | 0.16 (0.95)
  Dyspnoea: Week 7: number analyzed (Participants) | 132 | 156
  Dyspnoea: Week 7 | 0.30 (0.93) | 0.25 (0.92)
  Dyspnoea: Week 8: number analyzed (Participants) | 124 | 157
  Dyspnoea: Week 8 | 0.35 (0.87) | 0.24 (0.96)
  Dyspnoea: Week 9: number analyzed (Participants) | 125 | 159
  Dyspnoea: Week 9 | 0.34 (0.89) | 0.17 (0.91)
  Dyspnoea: Week 10: number analyzed (Participants) | 120 | 152
  Dyspnoea: Week 10 | 0.46 (0.93) | 0.16 (0.92)
  Dyspnoea: Week 11: number analyzed (Participants) | 117 | 156
  Dyspnoea: Week 11 | 0.39 (1.01) | 0.26 (0.96)
  Dyspnoea: Week 12: number analyzed (Participants) | 116 | 142
  Dyspnoea: Week 12 | 0.38 (0.96) | 0.22 (0.90)
  Dyspnoea: Week 13: number analyzed (Participants) | 108 | 142
  Dyspnoea: Week 13 | 0.34 (0.96) | 0.30 (1.02)
  Dyspnoea: Week 14: number analyzed (Participants) | 103 | 132
  Dyspnoea: Week 14 | 0.44 (0.95) | 0.22 (0.99)
  Dyspnoea: Week 15: number analyzed (Participants) | 101 | 133
  Dyspnoea: Week 15 | 0.45 (0.94) | 0.19 (0.95)
  Dyspnoea: Week 16: number analyzed (Participants) | 100 | 133
  Dyspnoea: Week 16 | 0.37 (1.06) | 0.26 (1.02)
  Dyspnoea: Week 17: number analyzed (Participants) | 97 | 131
  Dyspnoea: Week 17 | 0.35 (1.04) | 0.15 (1.00)
  Dyspnoea: Week 18: number analyzed (Participants) | 88 | 121
  Dyspnoea: Week 18 | 0.35 (0.99) | 0.22 (0.99)
  Dyspnoea: Week 19: number analyzed (Participants) | 81 | 122
  Dyspnoea: Week 19 | 0.30 (1.02) | 0.22 (0.97)
  Dyspnoea: Week 20: number analyzed (Participants) | 71 | 112
  Dyspnoea: Week 20 | 0.30 (1.09) | 0.27 (1.06)
  Dyspnoea: Week 21: number analyzed (Participants) | 74 | 114
  Dyspnoea: Week 21 | 0.22 (1.03) | 0.22 (1.05)
  Dyspnoea: Week 22: number analyzed (Participants) | 65 | 106
  Dyspnoea: Week 22 | 0.16 (1.10) | 0.28 (1.03)
  Dyspnoea: Week 23: number analyzed (Participants) | 65 | 106
  Dyspnoea: Week 23 | 0.24 (1.05) | 0.22 (1.03)
  Dyspnoea: Week 24: number analyzed (Participants) | 64 | 106
  Dyspnoea: Week 24 | 0.30 (0.98) | 0.24 (0.99)
  Dyspnoea: Week 25: number analyzed (Participants) | 60 | 100
  Dyspnoea: Week 25 | 0.50 (1.05) | 0.28 (0.99)
  Dyspnoea: Week 26: number analyzed (Participants) | 55 | 100
  Dyspnoea: Week 26 | 0.30 (1.05) | 0.24 (1.04)
  Dyspnoea: Week 27: number analyzed (Participants) | 55 | 99
  Dyspnoea: Week 27 | 0.43 (1.17) | 0.24 (1.06)
  Dyspnoea: Week 28: number analyzed (Participants) | 55 | 96
  Dyspnoea: Week 28 | 0.46 (1.02) | 0.25 (0.97)
  Dyspnoea: Week 29: number analyzed (Participants) | 54 | 99
  Dyspnoea: Week 29 | 0.43 (1.06) | 0.20 (1.01)
  Dyspnoea: Week 30: number analyzed (Participants) | 52 | 95
  Dyspnoea: Week 30 | 0.45 (1.08) | 0.21 (0.99)
  Dyspnoea: Week 31: number analyzed (Participants) | 44 | 93
  Dyspnoea: Week 31 | 0.35 (1.03) | 0.15 (0.99)
  Dyspnoea: Week 32: number analyzed (Participants) | 39 | 94
  Dyspnoea: Week 32 | 0.48 (1.03) | 0.16 (1.01)
  Dyspnoea: Week 33: number analyzed (Participants) | 41 | 85
  Dyspnoea: Week 33 | 0.36 (0.96) | 0.17 (0.95)
  Dyspnoea: Week 34: number analyzed (Participants) | 40 | 84
  Dyspnoea: Week 34 | 0.47 (1.15) | 0.24 (1.04)
  Dyspnoea: Week 35: number analyzed (Participants) | 39 | 87
  Dyspnoea: Week 35 | 0.42 (1.00) | 0.23 (1.03)
  Dyspnoea: Week 36: number analyzed (Participants) | 34 | 86
  Dyspnoea: Week 36 | 0.59 (1.06) | 0.22 (1.02)
  Dyspnoea: Week 37: number analyzed (Participants) | 33 | 86
  Dyspnoea: Week 37 | 0.53 (1.17) | 0.24 (1.03)
  Dyspnoea: Week 38: number analyzed (Participants) | 30 | 80
  Dyspnoea: Week 38 | 0.59 (1.06) | 0.22 (1.07)
  Dyspnoea: Week 39: number analyzed (Participants) | 32 | 72
  Dyspnoea: Week 39 | 0.65 (1.04) | 0.19 (1.01)
  Dyspnoea: Week 40: number analyzed (Participants) | 31 | 77
  Dyspnoea: Week 40 | 0.62 (1.02) | 0.19 (0.95)
  Dyspnoea: Week 41: number analyzed (Participants) | 30 | 74
  Dyspnoea: Week 41 | 0.63 (1.01) | 0.16 (0.95)
  Dyspnoea: Week 42: number analyzed (Participants) | 27 | 73
  Dyspnoea: Week 42 | 0.50 (1.01) | 0.17 (0.92)
  Dyspnoea: Week 43: number analyzed (Participants) | 23 | 76
  Dyspnoea: Week 43 | 0.32 (0.89) | 0.22 (0.90)
  Dyspnoea: Week 44: number analyzed (Participants) | 25 | 72
  Dyspnoea: Week 44 | 0.58 (0.83) | 0.23 (0.92)
  Dyspnoea: Week 45: number analyzed (Participants) | 25 | 69
  Dyspnoea: Week 45 | 0.49 (0.96) | 0.21 (0.90)
  Dyspnoea: Week 46: number analyzed (Participants) | 24 | 67
  Dyspnoea: Week 46 | 0.55 (1.02) | 0.23 (0.89)
  Dyspnoea: Week 47: number analyzed (Participants) | 23 | 63
  Dyspnoea: Week 47 | 0.53 (1.09) | 0.14 (0.90)
  Dyspnoea: Week 48: number analyzed (Participants) | 25 | 64
  Dyspnoea: Week 48 | 0.55 (0.96) | 0.14 (0.85)
  Dyspnoea: Week 49: number analyzed (Participants) | 23 | 62
  Dyspnoea: Week 49 | 0.63 (1.04) | 0.16 (0.90)
  Dyspnoea: Week 50: number analyzed (Participants) | 23 | 58
  Dyspnoea: Week 50 | 0.52 (0.98) | 0.24 (0.94)
  Dyspnoea: Week 51: number analyzed (Participants) | 21 | 62
  Dyspnoea: Week 51 | 0.67 (1.04) | 0.30 (0.97)
  Dyspnoea: Week 52: number analyzed (Participants) | 21 | 55
  Dyspnoea: Week 52 | 0.72 (1.02) | 0.27 (1.02)
  Dyspnoea: Week 53: number analyzed (Participants) | 23 | 54
  Dyspnoea: Week 53 | 0.81 (1.06) | 0.22 (0.95)
  Dyspnoea: Week 54: number analyzed (Participants) | 22 | 54
  Dyspnoea: Week 54 | 0.82 (1.06) | 0.23 (0.95)
  Dyspnoea: Week 55: number analyzed (Participants) | 21 | 49
  Dyspnoea: Week 55 | 0.77 (1.17) | 0.16 (0.99)
  Dyspnoea: Week 56: number analyzed (Participants) | 20 | 53
  Dyspnoea: Week 56 | 0.84 (1.15) | 0.18 (0.95)
  Dyspnoea: Week 57: number analyzed (Participants) | 17 | 46
  Dyspnoea: Week 57 | 0.68 (1.16) | 0.11 (0.91)
  Dyspnoea: Week 58: number analyzed (Participants) | 15 | 43
  Dyspnoea: Week 58 | 0.77 (1.06) | 0.16 (0.86)
  Dyspnoea: Week 59: number analyzed (Participants) | 13 | 40
  Dyspnoea: Week 59 | 0.66 (0.90) | 0.07 (0.85)
  Dyspnoea: Week 60: number analyzed (Participants) | 11 | 41
  Dyspnoea: Week 60 | 0.73 (0.96) | 0.27 (0.94)
  Dyspnoea: Week 61: number analyzed (Participants) | 13 | 43
  Dyspnoea: Week 61 | 0.85 (1.04) | 0.23 (0.90)
  Dyspnoea: Week 62: number analyzed (Participants) | 13 | 37
  Dyspnoea: Week 62 | 0.95 (1.05) | 0.16 (0.92)
  Dyspnoea: Week 63: number analyzed (Participants) | 12 | 36
  Dyspnoea: Week 63 | 0.67 (1.01) | 0.27 (0.95)
  Dyspnoea: Week 64: number analyzed (Participants) | 10 | 35
  Dyspnoea: Week 64 | 0.46 (0.78) | 0.14 (0.93)
  Dyspnoea: Week 65: number analyzed (Participants) | 9 | 33
  Dyspnoea: Week 65 | 0.40 (0.66) | 0.12 (0.95)
  Dyspnoea: Week 66: number analyzed (Participants) | 6 | 34
  Dyspnoea: Week 66 | 0.67 (0.74) | 0.16 (0.94)
  Dyspnoea: Week 67: number analyzed (Participants) | 7 | 30
  Dyspnoea: Week 67 | 0.37 (0.76) | 0.26 (1.01)
  Dyspnoea: Week 68: number analyzed (Participants) | 6 | 30
  Dyspnoea: Week 68 | 0.47 (0.80) | 0.25 (1.03)
  Dyspnoea: Week 69: number analyzed (Participants) | 7 | 29
  Dyspnoea: Week 69 | 0.43 (0.80) | 0.16 (1.11)
  Dyspnoea: Week 70: number analyzed (Participants) | 6 | 30
  Dyspnoea: Week 70 | 0.33 (0.83) | 0.07 (0.89)
  Dyspnoea: Week 71: number analyzed (Participants) | 5 | 26
  Dyspnoea: Week 71 | 0.40 (0.91) | 0.13 (0.89)
  Dyspnoea: Week 72: number analyzed (Participants) | 4 | 25
  Dyspnoea: Week 72 | -0.05 (0.25) | 0.06 (0.91)
  Dyspnoea: Week 73: number analyzed (Participants) | 4 | 24
  Dyspnoea: Week 73 | 0.45 (1.04) | 0.09 (0.99)
  Dyspnoea: Week 74: number analyzed (Participants) | 4 | 23
  Dyspnoea: Week 74 | 0.50 (1.01) | 0.27 (1.19)
  Dyspnoea: Week 75: number analyzed (Participants) | 4 | 21
  Dyspnoea: Week 75 | 0.55 (0.97) | 0.45 (1.31)
  Dyspnoea: Week 76: number analyzed (Participants) | 3 | 17
  Dyspnoea: Week 76 | -0.07 (0.12) | 0.02 (1.10)
  Dyspnoea: Week 77: number analyzed (Participants) | 2 | 17
  Dyspnoea: Week 77 | 0.00 (0.00) | 0.09 (1.17)
  Dyspnoea: Week 78: number analyzed (Participants) | 2 | 14
  Dyspnoea: Week 78 | 0.00 (0.00) | 0.03 (1.19)
  Dyspnoea: Week 79: number analyzed (Participants) | 2 | 14
  Dyspnoea: Week 79 | 0.00 (0.00) | 0.19 (1.18)
  Dyspnoea: Week 80: number analyzed (Participants) | 2 | 13
  Dyspnoea: Week 80 | 0.10 (0.14) | -0.26 (0.80)
  Dyspnoea: Week 81: number analyzed (Participants) | 2 | 12
  Dyspnoea: Week 81 | 0.10 (0.14) | -0.17 (1.15)
  Dyspnoea: Week 82: number analyzed (Participants) | 2 | 9
  Dyspnoea: Week 82 | 0.00 (0.00) | 0.18 (1.54)
  Dyspnoea: Week 83: number analyzed (Participants) | 2 | 4
  Dyspnoea: Week 83 | 0.00 (0.00) | 0.45 (1.22)
  Dyspnoea: Week 84: number analyzed (Participants) | 2 | 5
  Dyspnoea: Week 84 | 0.00 (0.00) | 0.60 (1.10)
  Dyspnoea: Week 85: number analyzed (Participants) | 1 | 5
  Dyspnoea: Week 85 | 0.20 (NA) — Only 1 participant. | 0.32 (1.53)
  Dyspnoea: Week 86: number analyzed (Participants) | 1 | 4
  Dyspnoea: Week 86 | 0.00 (NA) — Only 1 participant. | -0.15 (0.34)
  Dyspnoea: Week 87: number analyzed (Participants) | 1 | 3
  Dyspnoea: Week 87 | 0.20 (NA) — Only 1 participant. | -0.47 (0.23)
  Dyspnoea: Week 88: number analyzed (Participants) | 1 | 4
  Dyspnoea: Week 88 | 0.20 (NA) — Only 1 participant. | -0.70 (0.20)
  Dyspnoea: Week 89: number analyzed (Participants) | 1 | 2
  Dyspnoea: Week 89 | 0.20 (NA) — Only 1 participant. | -0.20 (0.57)
  Dyspnoea: Week 90: number analyzed (Participants) | 1 | 2
  Dyspnoea: Week 90 | 0.20 (NA) — Only 1 participant. | -0.50 (0.14)
  Dyspnoea: Week 91: number analyzed (Participants) | 1 | 2
  Dyspnoea: Week 91 | 0.00 (NA) — Only 1 participant. | -0.50 (0.14)
  Dyspnoea: Week 92: number analyzed (Participants) | 0 | 2
  Dyspnoea: Week 92 |  | -0.70 (0.14)
  Dyspnoea: Week 93: number analyzed (Participants) | 0 | 2
  Dyspnoea: Week 93 |  | -0.40 (0.28)
  Dyspnoea: Week 94: number analyzed (Participants) | 0 | 1
  Dyspnoea: Week 94 |  | -0.80 (NA) — Only 1 participant.
  Dyspnoea: Week 95: number analyzed (Participants) | 0 | 1
  Dyspnoea: Week 95 |  | -1.00 (NA) — Only 1 participant.
  Dyspnoea: Time of First Pd: number analyzed (Participants) | 110 | 96
  Dyspnoea: Time of First Pd | 0.58 (0.99) | 0.40 (1.06)
  Dyspnoea: Time of Last Tx Dose: number analyzed (Participants) | 141 | 150
  Dyspnoea: Time of Last Tx Dose | 0.47 (0.95) | 0.18 (0.94)

10. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Description: Minimum observed serum atezolizumab concentration (Cmin) prior to infusion at selected cycles (Arm A)
Time Frame: Predose (Prd; 0 hour [h]) on D1 of Cy 2,3,4,8,16 (Cy length=21 days) and thereafter on D1 of every 8th cycle (up to approximately 25 months)
Population: PK analyses were based on PK observations from all patients who received atezolizumab, carboplatin, cisplatin or pemetrexed treatment and who provided at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 247
μg/mL
  Cy2D1 | 69.8 (32.3)
  Cy3D1: number analyzed (Participants) | 228
  Cy3D1 | 115 (51.5)
  Cy4D1: number analyzed (Participants) | 213
  Cy4D1 | 151 (69.9)
  Cy8D1: number analyzed (Participants) | 145
  Cy8D1 | 221 (101)
  Cy16D1: number analyzed (Participants) | 76
  Cy16D1 | 234 (86.7)
  Cy24D1: number analyzed (Participants) | 13
  Cy24D1 | 257 (95.1)
  Treatment Discontinuation Visit: number analyzed (Participants) | 131
  Treatment Discontinuation Visit | 129 (93.1)
  Day 120 Post Last Dose: number analyzed (Participants) | 55
  Day 120 Post Last Dose | 13.4 (19.4)

11. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Description: Maximum observed serum atezolizumab concentration (Cmax) after infusion (Arm A)
Time Frame: Day 1 of Cycle 1 (Cycle length=21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 273
μg/mL | 403 (118)

12. Secondary Outcome: Plasma Concentrations for Carboplatin in Arm A(Atezolizumab + Carboplatin or Cisplatin + Pemetrexed)
Time Frame: Prd (0 h), 5-10 minutes (mins) before end of carboplatin infusion (infusion duration=1-2 h), 1 h post-infusion on D1 of Cy1,3 (Cy length=21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 27
ng/mL
  Cy1D1 Predose: number analyzed (Participants) | 24
  Cy1D1 Predose | NA (NA) — Predose of Cycle 1 Day 1 administration of Carboplatin.
  Cy1D1 Before End of Infusion: number analyzed (Participants) | 18
  Cy1D1 Before End of Infusion | 14900 (4260)
  Cy1D1 Post Infusion: number analyzed (Participants) | 23
  Cy1D1 Post Infusion | 12800 (4470)
  Cy3D1 Predose: number analyzed (Participants) | 20
  Cy3D1 Predose | 220 (83.8)
  Cy3D1 Before End of Infusion: number analyzed (Participants) | 17
  Cy3D1 Before End of Infusion | 17900 (4390)
  Cy3D1 Post Infusion: number analyzed (Participants) | 15
  Cy3D1 Post Infusion | 13900 (4080)

13. Secondary Outcome: Plasma Concentrations for Cisplatin in Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed)
Time Frame: Prd (0 h), 5-10 mins before end of cisplatin infusion (infusion duration=30-60 mins), 1 h post-infusion on D1 of Cy1,3 (Cy length=21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 10
ng/mL
  Cy1D1 Predose: number analyzed (Participants) | 9
  Cy1D1 Predose | NA (NA) — Predose of Cycle 1 Day 1 administration of Cisplatin.
  Cy1D1 Before End of Infusion: number analyzed (Participants) | 6
  Cy1D1 Before End of Infusion | 3630 (589)
  Cy1D1 Post Infusion: number analyzed (Participants) | 7
  Cy1D1 Post Infusion | 2400 (360)
  Cy3D1 Predose: number analyzed (Participants) | 8
  Cy3D1 Predose | 290 (86.1)
  Cy3D1 Before End of Infusion: number analyzed (Participants) | 7
  Cy3D1 Before End of Infusion | 3020 (968)
  Cy3D1 Post Infusion: number analyzed (Participants) | 7
  Cy3D1 Post Infusion | 2740 (543)

14. Secondary Outcome: Plasma Concentrations for Pemetrexed in Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed)
Time Frame: Prd (0 h), 5-10 mins before end of pemetrexed infusion (infusion duration=10 mins), 1 h post-infusion on D1 of Cy1,3 (Cy length=21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 36
ng/mL
  Cy1D1 Predose: number analyzed (Participants) | 34
  Cy1D1 Predose | NA (NA) — Predose of Cycle 1 Day 1 administration of Pemetrexed.
  Cy1D1 Before End of Infusion: number analyzed (Participants) | 26
  Cy1D1 Before End of Infusion | 86500 (41600)
  Cy1D1 Post Infusion: number analyzed (Participants) | 33
  Cy1D1 Post Infusion | 43600 (15800)
  Cy3D1 Predose: number analyzed (Participants) | 28
  Cy3D1 Predose | 1.83 (0.681)
  Cy3D1 Before End of Inufsion: number analyzed (Participants) | 22
  Cy3D1 Before End of Inufsion | 79400 (44400)
  Cy3D1 Post Infusion: number analyzed (Participants) | 27
  Cy3D1 Post Infusion | 50100 (26100)

15. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) of Atezolizumab
Description: Baseline prevalence and post-baseline incidence of anti-drug antibodies (ADA) to Atezolizumab in the Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed)
Time Frame: Prd (0 h) on D1 of Cy1,2,3,4,8,16 (Cy length=21 days) and thereafter on D1 of every 8th cycle, at treatment discontinuation & then every 30 days (up to 120 days) after last dose of atezolizumab (up to app 25 months)
Population: The ADA evaluable population was defined as patients with a non-missing baseline ADA sample and >=1 non-missing post-baseline ADA sample.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
Number analyzed (Participants) | 291
Percentage of Participants
  Baseline Evaluable Participants: number analyzed (Participants) | 277
  Baseline Evaluable Participants | 1.8
  Post-Baseline Evaluable Participants: number analyzed (Participants) | 271
  Post-Baseline Evaluable Participants | 35.4

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 13 December 2022 (up to approximately 80 months).
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any component of study treatment.
Groups:
- Arm B (Carboplatin or Cisplatin + Pemetrexed): Participants received IV infusion of 500 mg/m^2 pemetrexed on Day 1 q3w, and as per investigator's choice of either IV infusion of carboplatin on Day 1 q3w with a dose calculated using 'Calvert formula' to obtain AUC =6 mg/mL/min or IV infusion of 75 mg/m^2 cisplatin q3w on Day 1 q3w, during induction dosing period for 4 or 6 cycles (Cycle length=21 days). Participants who do not experience disease progression during the induction phase will begin maintenance therapy. Participants will receive IV infusion of 500 mg/m^2 of pemetrexed on Day 1 q3w until disease progression in the maintenance period.
Arm/Group | Arm B (Carboplatin or Cisplatin + Pemetrexed) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed
All-Cause Mortality (participants affected / at risk) | 189/286 | 190/292
Serious Adverse Events (participants affected / at risk) | 91/274 | 149/291
Other Adverse Events (participants affected / at risk) | 255/274 | 275/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B (Carboplatin or Cisplatin + Pemetrexed) (N=274) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed (N=291)
ANAEMIA (Blood and lymphatic system disorders) | 7 (10) | 11 (14)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 12 (12)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
PANCYTOPENIA (Blood and lymphatic system disorders) | 4 (6) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 11 (15)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (3) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 1 (1)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 4 (4)
AUTOIMMUNE COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 9 (9)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (2)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (3)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 6 (6)
ASTHENIA (General disorders) | 2 (2) | 5 (5)
CHEST PAIN (General disorders) | 2 (2) | 0 (0)
DEATH (General disorders) | 1 (1) | 2 (2)
DISEASE SUSCEPTIBILITY (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 2 (2)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 3 (4)
INFLAMMATION (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 2 (2) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 0 (0)
PAIN (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 2 (3) | 12 (12)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 2 (2)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 2 (2)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 3 (3)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
H3N2 INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
PERIPHERAL NERVE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 16 (17) | 17 (18)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 6 (9)
SEPSIS (Infections and infestations) | 2 (2) | 4 (4)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
TRACHEITIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 6 (6)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
STAB WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 3 (3)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (5) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 3 (3) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FRACTURE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HISTIOCYTIC NECROTISING LYMPHADENITIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR EMBOLISM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 1 (2)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 4 (4)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
DEVICE MALFUNCTION (Product Issues) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CATATONIA (Psychiatric disorders) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 3 (3)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (2) | 0 (0)
GLYCOSURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHRITIS ALLERGIC (Renal and urinary disorders) | 0 (0) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 2 (2)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
AORTIC EMBOLUS (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 1 (2) | 0 (0)
CONGESTIVE HEPATOPATHY (Hepatobiliary disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 0 (0) | 1 (1)
LARYNGOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Infections and infestations) | 1 (1) | 2 (2)
VASCULAR ACCESS SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CHANGE IN SEIZURE PRESENTATION (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm B (Carboplatin or Cisplatin + Pemetrexed) (N=274) | Arm A (Atezolizumab + Carboplatin or Cisplatin + Pemetrexed (N=291)
ANAEMIA (Blood and lymphatic system disorders) | 113 (142) | 129 (186)
NEUTROPENIA (Blood and lymphatic system disorders) | 38 (65) | 48 (95)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 23 (37) | 39 (60)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 18 (19)
LACRIMATION INCREASED (Eye disorders) | 18 (21) | 16 (16)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (7) | 15 (20)
CONSTIPATION (Gastrointestinal disorders) | 79 (96) | 92 (104)
DIARRHOEA (Gastrointestinal disorders) | 47 (56) | 60 (88)
DYSPEPSIA (Gastrointestinal disorders) | 9 (10) | 16 (18)
NAUSEA (Gastrointestinal disorders) | 114 (206) | 112 (266)
STOMATITIS (Gastrointestinal disorders) | 23 (26) | 35 (45)
VOMITING (Gastrointestinal disorders) | 49 (64) | 58 (81)
ASTHENIA (General disorders) | 54 (81) | 79 (118)
CHEST PAIN (General disorders) | 18 (18) | 22 (25)
FATIGUE (General disorders) | 68 (98) | 71 (116)
MALAISE (General disorders) | 17 (23) | 14 (23)
MUCOSAL INFLAMMATION (General disorders) | 19 (28) | 23 (24)
OEDEMA PERIPHERAL (General disorders) | 33 (38) | 46 (66)
PYREXIA (General disorders) | 37 (50) | 59 (89)
CONJUNCTIVITIS (Infections and infestations) | 15 (18) | 18 (23)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (13) | 16 (22)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 23 (29) | 52 (74)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 27 (35) | 51 (78)
BLOOD CREATININE INCREASED (Investigations) | 20 (26) | 34 (43)
NEUTROPHIL COUNT DECREASED (Investigations) | 48 (108) | 45 (116)
PLATELET COUNT DECREASED (Investigations) | 38 (69) | 38 (63)
WEIGHT DECREASED (Investigations) | 16 (17) | 26 (26)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 29 (67) | 20 (58)
DECREASED APPETITE (Metabolism and nutrition disorders) | 64 (84) | 78 (101)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 17 (20) | 15 (17)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 21 (29)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 14 (19) | 19 (31)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 (29) | 46 (61)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 25 (28) | 40 (51)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13 (13) | 23 (23)
DIZZINESS (Nervous system disorders) | 24 (27) | 19 (23)
DYSGEUSIA (Nervous system disorders) | 19 (19) | 28 (33)
HEADACHE (Nervous system disorders) | 24 (26) | 35 (39)
PARAESTHESIA (Nervous system disorders) | 14 (16) | 12 (13)
INSOMNIA (Psychiatric disorders) | 18 (18) | 28 (35)
COUGH (Respiratory, thoracic and mediastinal disorders) | 30 (36) | 43 (58)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 40 (42) | 44 (50)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 13 (16)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 17 (24) | 16 (35)
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 (7) | 20 (23)
PRURITUS (Skin and subcutaneous tissue disorders) | 16 (17) | 29 (37)
RASH (Skin and subcutaneous tissue disorders) | 21 (23) | 41 (54)
HYPERTENSION (Vascular disorders) | 7 (9) | 17 (31)
NASOPHARYNGITIS (Infections and infestations) | 8 (10) | 15 (20)
PNEUMONIA (Infections and infestations) | 11 (12) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02657434/Prot_002.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02657434/SAP_001.pdf